## **Reporting and Analysis Plan**

**Study ID: 208436** 

**Official Title of Study:** Reporting and Analysis Plan for a randomised, double-blind (sponsor unblinded), placebo-controlled, first time in human study to evaluate the safety, tolerability and pharmacokinetics of single (in both fed and fasted states) and repeat doses of GSK3186899 in healthy participants

Date of Document: 21-Nov-2019



# **GSK Vaccines Controlled Document**

 $\textbf{Documentum Name:} \quad \textbf{GSK3186899-208436 Statistical Analysis Plan Reporting and Analysis Plan Version 001}$ 

(18-Nov-2019)

Documentum Id: 090f45f689e7c46d

**Documentum Version:** 1.4

| Date (UTC date) | Signed by |
|-------------------------|------------------|
| 19-Nov-2019 10:47:00 AM | PPD |
| Justification | Sign as Approver |
| 21-Nov-2019 10:29:17 AM | PPD |
| Justification | Sign as Approver |
| Justification | |
| Justification | |
| Justification | |
| Justification | |
| Justification | |
| Justification | |
| Justification | |
| Justification | |



# **GSK Vaccines Controlled Document**

 $\textbf{Documentum Name:} \quad \textbf{GSK3186899-208436 Statistical Analysis Plan Reporting and Analysis Plan Version 001}$ 

(18-Nov-2019)

Documentum Id: 090f45f689e7c46d

**Documentum Version:** 1.4

| Date (UTC date) | Signed by |
|-----------------|-----------|
| Justification | |

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for a randomised, double-blind (sponsor unblinded), placebo-controlled, first time in human study to evaluate the safety, tolerability and pharmacokinetics of single (in both fed and fasted states) and repeat doses of GSK3186899 in healthy participants |
| <b>Compound Number</b> | : | GSK3186899 |
| Effective Date | : | [15-NOV-2019] |

## **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208436, which is a first time in human (FTiH) study comprising of a single and repeat ascending dose regimens in healthy participants, incorporating a food effect component.
- The key objective is to describe the safety, tolerability and pharmacokinetics of GSK3186899. Results from this study will also be used to identify appropriate and well tolerated doses of GSK3186899 and to investigate the influence of food on the PK of GSK3186899.
- This full RAP will be provided to the study team members to convey the content of the reporting efforts planned for the study informal interim analysis and final analysis deliverables for the Statistical Analysis Complete (SAC).
- All sections of the RAP have been populated in this version.

# Author(s)

| Author | Date |
|---|---|
| PPD | 15-Nov-2019 |
| Study Statisticia | |
| PPD | 16-Oct-2019 |
| Clinical Pharmacokineticist (Scientific Director, | |
| Quantitative Clinical Development (QCD), PAREXEL International) | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Review Confirmations (Method: E-mail)**

| Reviewer | Date |
|---|---|
| Project Statistician (Principal Statistician, FPD Clinical | 12-Nov-2019 |
| Statistics) PPD | |
| Operational Study Lead and Clinical Investigation Lead (Clinical Development Manager, R&D PCPS GCDO Clinical Unit Cambridge) | 16-Oct-2019 |
| PPD | |
| Medical Monitor (Head NCD Open Lab and Global Health Futures) | 16-Oct-2019 |
| PPD | |
| Safety and Medical Governance (SMG) Pharma Safety (formerly GCSP) representative (SERM Director, SMG Pharma Safety) 16-Oct-2019 | |
| PPD | 16-Oct-2019 |
| DQL (Principal Clinical Data Manager, R&D PCPS GCDO DM FPD) | |
| PPD | |
| Clinical Pharmacokineticist (Scientific Director Quantitative Clinical Development (QCD), PAREXEL International) 16-Oct-2019 | |
| PPD | |
| Study Programmer (Principal Programmer, FPD Clinical Statistics) | 16-Oct-2019 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| Diseases of the Developing World (DDW) Statistical Lead (Statistics Director, FPD Clinical Statistics) | To be updated after esigning is completed |
| Lead Programmers Line Manager (Programming Manager, FPD Clinical Programming) | To be updated after esigning is completed |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | ON | 8 |
| 2. | SLIMI | AARY OF | KEY PROTOCOL INFORMATION | 8 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | • | Objective(s) and Endpoint(s) | |
| | 2.3. | | Design | |
| | 2.4. | | cal Analyses | |
| 3. | DI AN | | ALYSES | 12 |
| J. | 3.1. | | Analyses | |
| | 0.1. | III(CIIIII | 3.1.1.1. Dose escalation meetings | 13 |
| | | | 3.1.1.2. Informal interim analysis | 14 |
| | | | 3.1.1.3. Safety review meetings | |
| | 3.2. | Final Ar | nalyses | |
| 4. | ΔΝΔΙ | VSIS PO | PULATIONS | 16 |
| ч. | 4.1. | | ol Deviations | |
| | 5.2. | | e Definitions | |
| | · | 5.2.1. | | |
| | 5.3. | Other C | Considerations for Data Analyses and Data Handling | |
| | | Conven | ntions | 21 |
| 6. | STUD | Y POPUI | LATION ANALYSES | 22 |
| | 6.1. | | ew of Planned Study Population Analyses | |
| 7. | CVEE | TV ANIAI | _YSES | 22 |
| ١. | 7.1. | | e Events Analyses | |
| | 7.2. | | e Events of Special Interest Analyses | |
| | 7.3. | | Laboratory Analyses | |
| | 7.4. | | Safety Analyses | |
| 8. | ДЦΛГ | | INICTIC ANALYSES | 24 |
| Ο. | 8.1. | | INETIC ANALYSEScal analyses of derived PK parameters | |
| | 0.1. | | Endpoints / Variables | |
| | | 0.1.1. | 8.1.1.1. Drug Concentration Measures | |
| | | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.2. | Summary Measure | <mark>26</mark> |
| | | 8.1.3. | Population of Interest | <mark>26</mark> |
| | | 8.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.1.5. | Statistical Analyses / Methods | |
| | 8.2. | Statistic part | cal analysis for comparison of food effect – Single dose stud | |
| | | 8.2.1. | Endpoints/Variables | |
| | | 8.2.2. | Summary Measure | |
| | | 8.2.3. | Population of Interest | |
| | | 8.2.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.2.5. | Statistical Analyses / Methods | 31 |
| | | | 8.2.5.1. Statistical Methodology Specification | 31 |

| | 8.3. | | al analysis for dose proportionality – Single and Repeat | |
|---|---|---|---|---|
| | | dose stu | dy parts | |
| | | 8.3.1. | Endpoints/Variables | |
| | | 8.3.2. | Summary Measure | |
| | | 8.3.3. | Population of Interest | |
| | | 8.3.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.3.5. | Statistical Analyses / Methods | |
| | | | 8.3.5.1. Statistical Methodology Specification | 35 |
| | 8.4. | Statistica | al analysis for dose accumulation – Repeat dose study part | 37 |
| | | 8.4.1. | Endpoints/Variables | 37 |
| | | 8.4.2. | Summary Measure | 37 |
| | | 8.4.3. | Population of Interest | |
| | | 8.4.4. | Strategy for Intercurrent (Post-Randomization) Events | 37 |
| | | 8.4.5. | Statistical Analyses / Methods | 39 |
| | | | 8.4.5.1. Statistical Methodology Specification | 39 |
| | 8.5. | Statistica | al analysis for time invariance ratio of GSK3186899 – | |
| | | Repeat of | dose study part | 41 |
| | | 8.5.1. | Endpoints/Variables | 41 |
| | | 8.5.2. | Summary Measure | 41 |
| | | 8.5.3. | Population of Interest | 41 |
| | | 8.5.4. | Strategy for Intercurrent (Post-Randomization) Events | 41 |
| | | 8.5.5. | Statistical Analyses / Methods | |
| | | | 8.5.5.1. Statistical Methodology Specification | 43 |
| 9. | REFE | RENCES. | | 45 |
| 40 | 4005 | NIDIOEO | | 40 |
| 10. | | | | 46 |
| | 10.1. | Appendi | x 1: Protocol Deviation Management and Definitions for Per | 40 |
| | | Protocol | Population | 46 |
| | 40.0 | 10.1.1. | Exclusions from Analysis Population | 46 |
| | 10.2. | | x 2: Schedule of Activities | 47 |
| | | 10.2.1. | Protocol Defined Schedule of Events in PART A (Cohorts 1-3) | 47 |
| | | 10.2.2. | Protocol Defined Schedule of Events in PART B (Cohorts | |
| | | | 4-6) | 50 |
| | 10.3. | Appendi | x 3: Assessment Windows | 56 |
| | | 10.3.1. | Definitions of Assessment Windows for Analyses | 56 |
| | 10.4. | Appendi | x 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | | 57 |
| | | 10.4.1. | Study Phases | 57 |
| | | | 10.4.1.1. Study Phases for Concomitant Medication | 57 |
| | | 10.4.2. | Treatment Emergent Flag for Adverse Events | 58 |
| | 10.5. | Appendi | x 5: Data Display Standards & Handling Conventions | 59 |
| | | 10.5.1. | Reporting Process | |
| | | 10.5.2. | Reporting Standards | |
| | | 10.5.3. | Reporting Standards for Pharmacokinetic | 60 |
| | 10.6. | Appendi | x 6: Derived and Transformed Data | |
| | | 10.6.1. | General | |
| | | 10.6.2. | Study Population | |
| | | 10.6.3. | Safety | |
| | | 10.6.4. | Pharmacokinetic | |
| | 10.7. | Appendi | x 7: Reporting Standards for Missing Data | 64 |

# CONFIDENTIAL

| | 10.7.1. | Premature Withdrawals | .64 |
|---|---|---|---|
| | 10.7.2. | Handling of Missing Data | .64 |
| | | 10.7.2.1. Handling of Missing and Partial Dates | |
| 10.8. | <b>Appendix</b> | 8: Values of Potential Clinical Importance | |
| | | Laboratory Values | |
| | | ECG | |
| | | Vital Signs | |
| 10.9. | <b>Appendix</b> | 9: Population Pharmacokinetic (PopPK) Analyses | .68 |
| 10.10. | Appendix | 10: Pharmacokinetic / Pharmacodynamic Analyses | .68 |
| 10.11. | Appendix | 11: Abbreviations & Trade Marks | .68 |
| | 10.11.1. | Abbreviations | .68 |
| | 10.11.2. | Trademarks | .70 |
| 10.12. | <b>Appendix</b> | 12: List of Data Displays | .71 |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Safety Tables | |
| | 10.12.6. | Pharmacokinetic Tables | .77 |
| | 10.12.7. | Pharmacokinetic Figures | .80 |
| | 10.12.8. | ICH Listings | .81 |
| | | Non-ICH Listings | |
| 10.13. | Appendix | : 13: Example Mock Shells for Data Displays | .89 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 208436:

| Protocol Revision Chronology: | | |
|---|---|---|
| Original Document Number: 2018N385133_00 | Dated: 09-JAN-2019 | Version: Original |
| Original Document Number: 2018N385133_01 | Dated: 19-MAR-2019 | Version: Amendment 01 |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no major changes or deviations to the originally planned statistical analysis specified in the Original Protocol 208436 (Dated: 09-Jan-2019) and the Amendment 01 (Dated: 19-Mar-2019).

A minor change is made to the first secondary objective where trough plasma concentration (Ctau) is removed from the SAD part and added to the MAD part after confirmation from the Study Pharmacokineticist.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the safety and tolerability of single and repeat doses of GSK3186899 in healthy participants | <ul> <li>Adverse event reporting, clinical laboratory safety data,<br/>physical examinations, vital signs, 12 lead ECGs, 24 hr<br/>telemetry</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the systemic pharmacokinetic (PK) profile of single (fasted and fed) and repeat doses of GSK3186899 in healthy participants | <ul> <li>Plasma concentrations of GSK3186899 plus derived parameters, as data allow.</li> <li>For SAD part: Derived PK parameters for GSK3186899 following single dose (fasted and fed) including area under the plasma drug concentration versus time curve (AUC(0-t), AUC(0-∞)), maximum observed plasma drug concentration (C<sub>max</sub>), time to maximum observed plasma drug concentration (T<sub>max</sub>), and apparent terminal half-life (T<sub>1/2</sub>) as data allow. Predicted accumulation Ratio (AR<sub>pred</sub>)# will be calculated.</li> <li>For MAD part: AUC(0-t), AUC(0-∞), AUC(0-tau), C<sub>max</sub>, trough plasma concentration (C<sub>tau</sub>), T<sub>max</sub> and T<sub>1/2</sub>.</li> </ul> |
| To examine dose proportionality<br>following single and multiple<br>doses of GSK3186899 | <ul> <li>Dose-proportionality assessment using derived PK parameters, as data allow:</li> <li>For SAD part: AUC(0-∞), C<sub>max</sub></li> </ul> |

| Objectives | Endpoints |
|---|---|
| | For MAD part: AUC(0-tau), C <sub>max</sub> , C <sub>tau</sub> |
| To assess accumulation and<br>time-invariance ratios of<br>GSK3186899 after multiple<br>doses | <ul> <li>Accumulation ratios assessment*, where data allow:<br/>RAUC(0-tau), RC<sub>max</sub>, RC<sub>tau</sub>. Time-invariance ratio<br/>calculation as AUC(0-12)<sup>†</sup> on day 10 to AUC(0-∞) on<br/>day 1.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To collect residual plasma<br>following GSK3186899 analysis,<br>and urine samples, for analysis<br>of metabolites of GSK3186899 | Metabolites of GSK3186899 in plasma and urine. These analyses will be detailed in a separate analysis plan. |
| To collect bile sample for<br>analysis of metabolites of<br>GSK3186899 (Part A fed<br>regimen only) | Metabolites of GSK3186899 in bile. These analyses will<br>be detailed in a separate analysis plan. |

<sup>\*</sup> Accumulation ratios calculated as the ratio of last dose to first dose PK parameters: RAUC<sub>(0-tau)</sub> = AUC<sub>(0-tau)</sub> on last dose to AUC<sub>(0-tau)</sub> on first dose, RCmax = Cmax on last dose to Cmax on first dose, RCtau = Ctau on last dose to Ctau on first dose. # ARpred = 1/(1-e^(k\*tau)) where k is elimination rate constant following the single dose and tau is the dosing interval for the intended repeat dosing.

<sup>†</sup> It is AUC(0-12) if dosing is BID, or, AUC(0-8) if dosing is TID.

# 2.3. Study Design



## Overview of Study Design and Key Features under fasted conditions and 1 regimen under fed conditions. The fed conditions regimen will investigate the safety, tolerability and PK of a single dose of GSK3186899 following food administration. Part B will be a twice-daily (BID) 10-day repeat dose design in up to 3 parallel cohorts of participants (Cohorts 4, 5 and 6). Part B may include drug administration after either fed or fasted conditions, this will be dependent on the interim results from Part A. If under fasted conditions, participants will be required to fast at least 2 hours before and after drug administration. Dosing Part A (single ascending dose) For Part A, the dose escalation phase, up to 3 cohorts may be used (Cohorts 1-3). Cohorts 1 and 2 will consist of 8 healthy participants each. If used, Cohort 3 will consist of up to 14 healthy participants. For Cohorts 1 and 2, each participant will receive a maximum of 3 ascending oral doses of GSK3186899 and 1 placebo dose under fasted conditions. At each dose level, GSK3186899 and placebo will be administered in a 3:1 ratio, within each period, according to the randomization schedule in a blinded manner. Up to a maximum of 7 dose levels will be studied in Part A as illustrated in Figure 1 above. For Cohort 3, each participant will receive 1 oral dose of GSK3186899 selected based on the results from Cohorts 1 and 2, under both fasted and fed conditions. For each cohort and within each treatment period (except Cohort 3), the first 2 participants will act as sentinels. No participant will be a sentinel participant more than once. On Day 1, 1 of the 2 sentinel participants will receive the active dose and the other will receive placebo. Based on the Principal Investigator's review of the 2 sentinel participants after at least the first 24hr post-dose safety data (e.g. vital signs, ECGs and AEs), the remaining 6 participants can then be randomized to dosing. Part B (repeat dose) For the repeat dose escalation phase in Part B, there will be up to 3 cohorts (Cohorts 4, 5 and 6), consisting of 8 healthy participants randomised to receive repeat doses of either GSK3186899 or placebo, administered in a 3:1 ratio according to the randomization schedule in a blinded manner. For BID dosing, GSK3186899 or placebo will be administered using a 12hr dosing interval. Based on emerging data in Part A, an alternate dosing regimen (OD or TID) may be selected if deemed suitable. The first 2 participants in each cohort in Part B will act as sentinels. On Day 1 • until Day 10, 1 of the 2 sentinel participants will receive the active dose twice daily and the other will receive placebo twice daily. Once these participants have completed their first 5-days of dosing, the safety and tolerability data will be reviewed by the Principal Investigator. If there are no clinically relevant safety or tolerability concerns (e.g. vital signs, ECGs and AEs) the remaining 6 participants will be randomized to dosing. Time & Refer to Appendix 2: Schedule of Activities **Events** Treatment Part A consists of up to 30 participants in up to 3 cohorts (excluding possible **Assignment** replacements): Cohort 1 and 2 will each have 6 participants in active versus 2 participants in placebo (i.e., in a 3:1 ratio)

| Overview of \$ | Study Design and Key Features |
|---|---|
| | <ul> <li>Cohort 3 will contain up to 14 participants in a 1:1 ratio for (fed and<br/>active) versus (fasted and active)</li> </ul> |
| | <ul> <li>Part B consists of up to 24 participants in up to 3 cohorts:</li> <li>Cohorts 4, 5 and 6 will each have 6 participants in active versus 2 participants in placebo (i.e., in a 3:1 ratio)</li> </ul> |
| Interim<br>Analysis | No formal interim analyses (IA) are planned for this study. However, safety, tolerability, and PK data will be reviewed before each dose escalation in Part A (single dose) and Part B (repeat dose), prior to the investigation of the food effect, and between Part A and Part B. An informal interim analysis for Part A will be conducted prior to initiating Part B. This analysis will support the decision to progress or not to progress to Part B. |

# 2.4. Statistical Analyses

Given that this is a FTiH study, statistical analyses planned will be mainly descriptive in nature involving frequencies and percentages for categorical variables and number of subjects (n), mean, standard deviation, median, minimum and maximum for continuous variables.

Where appropriate (for e.g., evaluation of dose proportionality, drug accumulation, food effect) statistical modelling will be performed and point estimates with 90% confidence intervals (CIs) will be constructed.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal interim analyses (IA) are planned for this study. However, regular dose escalation meetings, an informal IA and safety review meetings are planned to be performed at different time points described below.

- Dose escalation meetings are planned to review the safety, tolerability, and PK data prior to:
  - o each dose escalation in Part A (single dose) Cohorts 1 and 2,
  - o initiation of the food effect Cohort 3, and
  - o each dose escalation in Part B (repeat dose) prior to initiation of Cohorts 5 and 6
- An informal IA to review the safety, tolerability, and PK data from Part A is planned prior to:
  - o progression to Part B.
- Additional instream safety review meetings including all safety and tolerability data only are planned prior to:
  - o progression to Cohort 2 in Part A
  - o progression to Period 2 in the food effect Cohort 3.

There will not be a formal database freeze performed for this informal IA. Data included for these analyses will be as complete and clean as possible based on continuous data review and monitoring activities.

The final study analysis post- database freeze will include all data captured in the study database.

## 3.1.1.1. Dose escalation meetings

Statistical displays will not be produced by Biostatistics for the dose escalation meetings. During the meeting, safety data (presented by the CUC Principal Investigator or delegate) and PK data (presented by Study Pharmacokineticist or delegate) will be reviewed by the committee.

The meeting will discuss blinded data in an open forum with the GSK Study team members and Principal Investigator (or their delegate) in attendance. If required, the data may be reviewed in an unblinded fashion by the unblinded members including the SMG (formally GCSP) Safety representative and Study Pharmacokineticist.

The decision to proceed to the next dose level of GSK3186899 will be made at a DEC meeting based on:

• all available safety and tolerability data from individuals (including AEs, laboratory safety tests, telemetry, ECGs and vital signs) from a minimum of 48 hours post-dose (10 days for repeat dose) from a minimum of 4 or more participants who have received GSK3186899 at the current dose level

• all available safety and tolerability data accumulated from preceding single/repeat dose levels and available PK data from current (minimum of 4 or more participants) and preceding single/repeat dose levels.

Further details of the DEC membership, data to be reviewed and stopping criteria are outlined in the DEC charter.

## 3.1.1.2. Informal interim analysis

An informal interim analysis (IA) after completion of Part A will be conducted prior to initiation of Part B. This analysis will support the decision to progress, or, not progress to Part B and will consist of the following statistical displays on blinded safety and blinded PK data. Safety tables will therefore be presented by period rather than treatment to maintain the blind of the study.

Table 1: Planned Statistical Displays for the Interim analysis

| SI.<br>No. | Population | IDSL /<br>Example<br>Shell | Title | Responsible function |
|---|---|---|---|---|
| 1 | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 2 | Safety | ES3 | Listing of Reasons for Study Withdrawal – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 3 | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 4 | Safety | DM3 | Summary of Demographic Characteristics – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 5 | Safety | DM4 | Listing of Demographic Characteristics - Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 6 | Safety | EX1 | Summary of Exposure to Study Treatment - Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 7 | Safety | EX4 | Listing of Exposure Data – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 8 | Safety | AE1CP | Summary of All Adverse Events by System<br>Organ Class and Preferred Term - Part A<br>(Cohort 1 and Cohort 2 only) | Biostatistics |
| 9 | Safety | AE9 | Listing of All Adverse Events - Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 10 | Safety | EG4 | Listing of All ECG Values for Subjects with<br>Any Value of Potential Clinical Importance -<br>Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 11 | Safety | EG6 | Listing of All ECG Findings for Subjects with<br>an Abnormal Finding - Part A (Cohort 1 and<br>Cohort 2 only) | Biostatistics |
| 12 | Safety | LB6 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical | Biostatistics |

| | | | Importance – Part A (Cohort 1 and Cohort 2 only) | |
|---|---|---|---|---|
| 13 | Safety | UR2B | Listing of All Urinalysis Data for Subjects with<br>Any Value of Potential Clinical Importance -<br>Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 14 | Safety | VS5 | Listing of All Vital Signs for Subjects with values Potential Clinical Importance - Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 15 | Safety | EG6 (to be modified for telemetry data) | Listing of Telemetry findings - Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 16 | Safety | DV2 | Listing of Important Protocol Deviations – Part A (Cohort 1 and Cohort 2 only) | Biostatistics |
| 17 | PK | Non<br>standard<br>shell | Summary of Untransformed Derived<br>GSK3186899 Plasma Pharmacokinetic<br>Parameters by dose and fed status - Part A<br>(All Cohorts) | CPMS |
| 18 | PK | Non<br>standard<br>shell | Summary of the ratio of fed versus fasted on AUC(0-∞) and Cmax – Part A Cohort 3 | CPMS |
| 19 | PK | Non<br>standard<br>shell | Geo Mean (+ SD) GSK3186899 Plasma<br>Concentration-Time Plot (Linear and Semi-<br>Log) – Part A (Cohort 1 and Cohort 2 only) | CPMS |
| 20 | PK | Non<br>standard<br>shell | Box Plot of AUC(0-∞) and Cmax versus dose (Linear) – Part A (Cohort 1 and Cohort 2 only) | CPMS |
| 21 | PK | Non<br>standard<br>shell | Box Plot of dose normalised AUC(0-∞) and Cmax versus dose (Linear) – Part A (Cohort 1 and Cohort 2 only) | CPMS |
| 22 | PK | Non<br>standard<br>shell | Geo Mean (+ SD) GSK3186899 Plasma<br>Concentration-Time Plot (Linear and Semi-<br>Log) grouped by fed and fasted status – Part<br>A Cohort 3 | CPMS |
| 23 | PK | Non<br>standard<br>shell | Box Plot of AUC (0-∞) and Cmax (Linear) grouped by fed and fasted status – Part A Cohort 3 | CPMS |
| 24 | PK | Non<br>standard<br>shell | Listing of GSK3186899 Plasma<br>Pharmacokinetic Concentrations (loge-<br>transformed) -Time Data by dose - Part A<br>(All Cohorts) | CPMS |

The PK related displays will be prepared by/under the auspices of the CPMS function and the safety related displays will be prepared by/under the auspices of the Biostatistics function.

The safety related IA displays will include data from Cohort 1 and Cohort 2 only. This is because all the doses will be investigated for safety and tolerability during these two cohorts and Cohort 3 will provide further information on the fed or fasted regimen to be applied in the Part B, for multiple ascending doses.

The actual treatment information will not be presented in any displays. Aggregated data will be reported in the tables of safety endpoints. The PK data will be presented without subject IDs. Blinded listings of safety and PK data will be provided.

A blinded dry run will be performed prior to the informal IA. The dry run displays will be reviewed by the study team including SMG Pharma Safety representative.

If required and/or requested by the DEC, an independent statistician and programmer(s) may be deployed to create unblinded displays.

However, a support pharmacokineticist in GSK will have access to extract scrambled PK data from SMS2000 to PKHARP and transfer the data via secured email to the Study pharmacokineticist (in PAREXEL International) for their reviews and analyses during study.

In case, there are any serious adverse events requiring further investigation, the unblinded SMG Pharma Safety representative and unblinded Study Pharmacokineticist can support further investigation.

# 3.1.1.3. Safety review meetings

The decision to proceed from Cohort 1 Period 4 to Cohort 2 Period 1 and similarly progress from Cohort 3 Period 1 (DLX) to Cohort 3 Period 2 (DLX-FD) will be made by the Principal Investigator and Medical Monitor based on all available safety and tolerability data from a minimum of 48 hours post-dose from a minimum of 4 or more participants who have received GSK3186899 at the current dose level. Individual safety data (AEs, laboratory safety tests, telemetry, ECGs and vital signs) will also be reviewed. PK data will not be included in these reviews.

The study team will remain blinded until the database freeze, except for the unblinded site Pharmacist, unblinded study Pharmacokineticist and SMG Pharma Safety representative.

# 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) have been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

A final blinded dry run will be performed prior to the database lock for review by the study team.

## 4. ANALYSIS POPULATIONS

For purposes of analysis, the following populations are defined:

| Population | Description | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Screen Failure |
| Enrolled | All participants who passed screening and entered the study. Included are: Randomized Participants | Study Population |
| | Note: screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | |
| Safety | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> Note: Participants who were not randomized but received at least | <ul><li>Study Population</li><li>Safety</li></ul> |
| | one dose of study treatment should be listed. | |
| PK | All participants in the Safety population who had at least 1 non-missing PK assessment* (Non-quantifiable [NQ] values will be considered as non-missing values). | • PK |

Refer to ****: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (PDs), including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [Version 1.0 dated 10 April 2019 or later].

Exclusion from the analysis sets due to a deviation will be determined programmatically using the criteria described in the table of Analysis populations above. These deviations will not be included in the SDTM dataset but will be programmed in the protocol deviation analysis (ADaM) dataset. This dataset will be the basis for the summaries and listings of protocol deviations.

Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

<sup>\*</sup> PK assessments refer to the plasma concentrations and not the PK parameters.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays f | or Reporting |
| Code | Description | Description | Order in TLF |
| | PART A | | |
| P1 / P2 | Placebo cohort 1 / Placebo cohort 2 | Placebo Part A | 1 |
| D1 | GSK3186899 Dose Level 1 | GSK 30 mg | 2 |
| D2 | GSK3186899 Dose Level 2 | GSK 60 mg | 3 |
| D3 | GSK3186899 Dose Level 3 | GSK 120 mg | 4 |
| D4 | GSK3186899 Dose Level 4 | GSK 300 mg | 5 |
| D5 | GSK3186899 Dose Level 5 | GSK 600 mg | 6 |
| D6 | GSK3186899 Dose Level 6 | GSK 800 mg | 7 |
| D7 | GSK3186899 Dose Level 7 | GSK X.X mg | 8 |
| | (this dose was not investigated) | | |
| DX-FA | GSK3186899 Dose Level X fasted | GSK X.X mg fasted | 9 |
| DX-FE | GSK3186899 Dose Level X fed | GSK X.X mg fed | 10 |
| | PART B | | |
| P4/ P5/ P6 | Placebo cohort 4/ Placebo cohort 5/<br>Placebo cohort 6 | Placebo Part B | 1 |
| R1 | GSK3186899 Repeat Dose Level 1 | GSK X.X mg BID | 2 |
| R2 | GSK3186899 Repeat Dose Level 2 GSK X.X mg BID 3 | | 3 |
| R3 | GSK3186899 Repeat Dose Level 3 | GSK X.X mg BID | 4 |

Note: Doses levels 1 to 6 were known at the time of RAP finalisation. The later doses were unknown, but will be known and detailed in the final study reporting.

For Part A, this order of the treatments will be considered for displays including all treatment groups from Cohorts 1, 2 and 3. However, for displays by Cohorts, only relevant treatment groups will be presented in the same ascending order mentioned above.

Treatment comparisons will be displayed using the descriptors as specified below:

- In general, comparison between 2 doses: GSK X.X mg vs GSK X.X mg
- In Cohort 3 (same dose different food regimen): GSK X.X mg fed vs fasted.

#### 5.2. Baseline Definitions

Baseline is defined as the last non-missing pre-dose assessment in each cohort. In general, assessments on Study day 1 taken prior to first dose are used as baseline. In some unlikely situations described below, the baseline will be defined as:

- when there are multiple assessments captured on Day 1, but the time of the first assessments is missing, then this first recorded assessment will be considered as the baseline
- when only one assessment is captured on Day 1 with time of assessment as
  missing, then conservatively the last available assessment from Day -1 or prior
  will be defined as the baseline
- when there are no assessments collected at Day 1, the last available data from either Day -1/ Day -2 or screening (as schedule of assessment in each Part/Cohort permits) will be defined as baseline
- when pre-dose data is completely missing for a subject, then no derivation will be performed, and the baseline will be set to missing

In Part A, for each period within a cohort, the period baseline is defined in a similar manner, by considering the last available non-missing pre-dose assessment in that period.

For some ECG and Vital Signs parameters, the pre-dose data is captured as triplicate. In these cases, the baseline will be defined as the mean of the assessments.

In addition, for some PK endpoint analyses, the adjusted baselines may be considered, if the pre-dose PK concentration value in a period is observed to be greater than 5% of the previous dose Cmax value:

- Subject level baseline is defined as the mean of baseline across periods for each subject. If a period baseline is missing, the mean of available period baselines will be considered as baseline.
- Period level baseline is defined as the difference between the baseline value and subject level baseline for each period and each subject.

## 5.2.1. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from baseline in the study | |
| Change from Baseline | = Post-dose visit value – Baseline value |
| % Change from Baseline | = 100 x [(Post-dose visit value – Baseline value) / Baseline value] |
| Change from baseline within a period | |
| Change from Baseline in Period X | = Period X Post-dose value – Period X baseline value |

| % Change from Baseline in Period X | = 100 x [(Period X Post-dose value – Period X baseline value) / Period X baseline value] |
|---|---|

## NOTES:

- O Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definitions (the baseline of the study and the baseline of each period (unadjusted)) will be used for derivations for endpoints / parameters and indicated on summaries. Unless otherwise stated, if baseline data is missing or post-dose data is missing no derivation will be performed and (%) change from baseline will be set to missing.
- The relevant baseline definition will be footnoted on all displays involving change from baseline.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Schedule of Activities |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. In this document, Appendix 12 contains a list of data displays and analysis sets planned for the informal interim analysis.

Details of the planned displays and analysis sets for final study reporting will be presented in ****: List of Data Displays.

## 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, consisting all subjects who had a dose (including those who had partial dose) of study treatment.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and common ( $\geq$  5%) AEs by overall frequency will be based on GSK Core Data Standards. The details of the planned displays are provided in ****: List of Data Displays.

# 7.2. Adverse Events of Special Interest Analyses

Adverse events of special interest are those considered possibly related to/associated with stomach erosion, adrenal insufficiency and renal impairment.

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of final reporting. The details of the planned displays are provided in ****: List of Data Displays.

# 7.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, Renal and Liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in ****: List of Data Displays.

# 7.4. Other Safety Analyses

The analyses of non-laboratory safety test results including vital signs, 12 lead ECG and 24-hour telemetry will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in ****: List of Data Displays.

# 8. PHARMACOKINETIC ANALYSES

All PK analyses planned for the study are a part of the secondary objectives.

## 8.1. Statistical analyses of derived PK parameters

## 8.1.1. Endpoints / Variables

## 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Standards for Pharmacokinetic).

## 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin version 8.0. All calculations of non-compartmental parameters will be based on actual sampling times.

For dose escalation meeting and interim analysis planned sampling times may be used if actual timepoints are not available.

Pharmacokinetic parameters listed will be determined from the plasma concentrationtime data, provided there is enough evaluable data available for the calculations. If the concentration data is available partially, then based on scientific judgement the data will be assessed for inclusion or exclusion from the analysis.

| Parameter | Parameter Description |
|---|---|
| Plasma PK Para | Plasma PK Parameters: |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| RCmax | Ratio of Cmax on last dose to Cmax on first dose, i.e., |
| | $RCmax = \frac{Cmax \ on \ the \ last \ dose}{Cmax \ on \ the \ first \ dose}.$ |
| Ctau | Trough concentration determined directly from the concentration data (only for Part B of the study). It will be the concentrations at 12h or 8h after first dose (if BID or TID administration, respectively) and always concentration at pre-dose on the last dose. |
| RCtau | Ratio of Ctau on last dose to Ctau on first dose, i.e., |
| | $RCtau = rac{Ctau \ on \ the \ last \ dose}{Ctau \ on \ the \ first \ dose}$ |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| tlag* | Lag time before first observation of drug concentrations (after single dose only) |

| Parameter | Parameter Description |
|---|---|
| Tlast* | Time of last quantifiable concentration |
| t <sub>1/2</sub> | Apparent terminal half-life will be calculated as: |
| | $t_{1/2} = \frac{\ln 2}{\lambda_n}$ |
| | $\lambda_{1/2} = \lambda_{z}$ |
| | (NOTE: $\lambda_z$ is the terminal phase rate constant). |
| AUC(0-24h) | Area under the concentration-time curve from time zero to 24 hours post-dose (after single dose only). |
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration $(C(t))$ will be calculated using the linear trapezoidal rule for each incremental trapezoid and the $\log_e$ trapezoidal rule for each decremental trapezoid. |
| AUC(0-tau) | Area under the concentration-time curve from time zero to the time of the trough concentration (C(tau)) will be calculated for Part 2 of the study only (repeat dose) using the linear trapezoidal rule for each incremental trapezoid. |
| RAUC(0-tau) | AUC(0-tau) on last dose to AUC(0-tau) on first dose |
| | $RAUC(0 - tau) = \frac{AUC(0 - tau) \text{ on the last dose}}{AUC(0 - tau) \text{ on the first dose}}$ |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated (after single dose only) as: |
| | $AUC(0-\infty) = AUC(0-t) + \frac{C(t)}{\lambda z}$ |
| | (NOTE: $\lambda z$ is the terminal phase rate constant. % of the extrapolated area should not exceed 20%. Any value of AUC(0- $\infty$ ) derived with more than 20% extrapolation should be flagged and excluded from summary statistics if >30%). |
| AR <sub>pred</sub> | AR <sub>pred</sub> is calculated as: |
| | $ARpred = \frac{1}{1 - e^{k*tau}}$ |
| | where k is elimination rate constant following the single dose and tau is the dosing interval for the intended repeat dosing. |
| R <sup>2</sup> adjusted* | The goodness of fit statistic for the terminal elimination phase, adjusted for the number of points used in the estimation of $\lambda z$ . |
| λΖ | $\lambda_z$ is the terminal phase rate constant. A minimum number of three data points in the terminal phase will be used starting at any post-Cmax data point. The adjusted correlation coefficient (R² adjusted) in general should be greater than 0.90. Any value < 0.90 but $\geq$ 0.8 will be flagged but may be used at the PK Scientist's best knowledge and judgment, any value <0.8 should be considered for exclusion from the statistical analysis. All the derived parameters that include $\lambda z$ in their calculation (i.e, t½, AUC(0- $\infty$ ) will need to be flagged or excluded from statistical analysis accordingly. The interval used to determine $\lambda z$ should be equal or greater than 1.5-fold the estimated half-life or otherwise flagged and used at the PK Scientist's best knowledge and judgment. |
| λz upper limit* | The upper limit on time for values to be included in the calculation of λz. |

| Parameter | Parameter Description |
|---|---|
| λz lower limit* | The lower limit on time for values to be included in the calculation of $\lambda z$ |
| λz number of points* | The number of time points used in computing λz. |
| % AUCex* | Percent of AUC <sub>∞</sub> that is extrapolated beyond last quantified concentration |
| CL/F* | The apparent clearance will be calculated only for Part 1 of the study (single dose) as Dose/ AUC(0-∞) |
| CLss* | The apparent clearance at steady state will be calculated only for day 10 Part 2 of the study (repeat dose) as Dose/ AUC(0-tau) |
| Urine PK Parameters: | |
| Ae <sub>(t1-tz)</sub> * | Amount excreted in the urine at each interval collection (24 h) |
| fe <sub>(0-tz)</sub> * | The fraction of unchanged drug excreted in urine will be calculated as $f_e = A_e/Dose$ , up to tz hours, where tz is the last collection time |
| CL <sub>R</sub> * | Renal Clearance calculated as Ae <sub>(0-tz)</sub> / AUC <sub>(0-tz)</sub> |

#### NOTES:

• \*Additional exploratory parameters have been included which will be listed only.

# 8.1.2. Summary Measure

All the derived PK parameters will be summarized descriptively.

Detail methods and displays of the summary measures are specified in Section 8.1.6 Statistical Analyses/ Methods.

Some of the parameters in the list above will be used for statistical modelling, as described in the subsequent analyses sections.

## 8.1.3. Population of Interest

These descriptive summaries will be based on the PK population.

## 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

In Table 2 below, the possible intercurrent events and the rationale for relating them to treatment or otherwise is described. Once a subject discontinues from study treatment, they will proceed straight to follow up and no further data will be collected.

Individual subject data will be included in data listings regardless of the strategies followed for the analyses.

If feasible, subjects will be replaced until the desired sample size is attained.

## **Table 2 Strategies for Intercurrent events**

| Intercurrent events | Relation to treatment and rationale | Strategy, rationale and details of action taken |
|---|---|---|
| Subject<br>withdraws<br>study<br>consent | Not related to treatment/ Subject drops out due to logistic reasons and not due to any event related to treatment | <ul> <li>The strategy will be a While-on-Treatment strategy, where we are interested in the treatment effects prior to the withdrawal only.</li> <li>Subjects' data available up to the withdrawal will be included in the descriptive PK summaries.</li> <li>If a subject withdraws consent during a period, the missing data post withdrawal will not be imputed.</li> <li>The derived PK parameters for e.g., AUC, C<sub>max</sub> etc. of that partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria).</li> </ul> |
| Subject does not take the full treatment | Not related to treatment/ The treatment will be administered as a powder dissolved in diluent. To ensure all treatment is ingested, the bottle containing the dispersion will be rinsed three times and the subject will be expected to ingest this in addition to the initial dispersion. If three rinses are not all ingested, the subject may not take the full treatment dose. | In the current formulation, it is hard to measure the exact proportion of dose ingested if not all rinses are taken. It is also uncertain whether the formulation could change in future development. To account for this, we propose two different strategies described below. If this intercurrent event is not observed, then both strategies will provide the same results and only the hypothetical strategy will be presented for the final analysis. Primary analysis - The strategy will be a Hypothetical strategy, where we are interested in the treatment effects in a hypothetical scenario where all subjects have taken complete dose. - In this case, the data from a period in which an incomplete dose is taken would be considered as missing at random and excluded from analyses. - If the drug formulation is changed in the future studies, this estimate will provide the true relationship between the actual dose intake and its exposure under this strategy. Supplementary analysis - The strategy will be a Treatment policy |

| | | - | treatment effects regardless of the actual amount of dose taken. The analysis will include PK parameters derived based on concentrations of both complete and partial doses (if data permits based on criteria described in Section 8.1.1.2) and will be analysed using the nominal or prescribed dose. If the drug formulation remains unchanged in the future studies, this estimate will provide the true relationship between a nominal dose and its exposure under this strategy, i.e., a close to real-world situation. |
|---|---|---|---|
| Subject<br>drops out<br>due to<br>Adverse<br>events | Related to treatment/ If the adverse event is confirmed to be related to study treatment | - | The primary strategy will be a <b>Hypothetical</b> strategy, where we are interested in the treatment effects in a hypothetical scenario where discontinuation due to an AE would not happen. The missing data after discontinuation will assumed to be missing at random The derived PK parameters of the last fully or partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |

## 8.1.5. Statistical Analyses / Methods

For parameters tabulated in Section 8.1.2, data will be summarized using the following descriptive statistics.

- N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum for the untransformed data
- Geometric mean, 95% CI for the geometric mean, SD of log<sub>e</sub>-transformed data and %CV<sub>b</sub> or %CVw for the untransformed data (except Tmax and T<sub>½</sub>)
- Based on the intercurrent events observed in the study, appropriate strategies from Table 2 in Section 8.1.4 will be considered for handling of missing data (if any) and interpretation of the analysis results. If multiple intercurrent events are observed (for e.g., if the subject does not take the full treatment as well he withdraws study consent), then the data will be handled using more than one strategy as described in Table 2 and interpretations of the results will be made accordingly.

Graphical presentations will be provided if appropriate. All data will be listed. Details of the planned displays are provided in ****: List of Data Displays and will be based on GSK Data Standards and statistical principles.

# 8.2. Statistical analysis for comparison of food effect – Single dose study part

# 8.2.1. Endpoints/Variables

To assess the food effect in Cohort 3, the statistical analysis will be based on AUC(0-t),  $AUC(0-\infty)$  and Cmax, only.

## 8.2.2. Summary Measure

The summary measure will be the point estimates and 90% CIs of mean differences of GSK3186899 fed – GSK3186899 fasted, based on the loge-transformed data, and after back-transformation of this estimated differences, the geometric mean ratios of (GSK3186899 fed: GSK3186899 fasted) will be presented.

## 8.2.3. Population of Interest

These analyses will be based on the PK population.

# 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

In the Table 3 below, the possible intercurrent events and the rationale for relating them to treatment or otherwise is described. Once a subject discontinues from study treatment, they will proceed straight to follow up and no further data will be collected.

All subjects' data will be included in data listings irrespective of the strategies followed for the analysis.

If feasible, subjects will be replaced until the desired sample size is attained.

**Table 3 Strategies for Intercurrent events** 

| Intercurrent events | Relation to treatment and rationale | Strategy, rationale and details of action taken |
|---|---|---|
| Subject<br>withdraws<br>study<br>consent | Not related to treatment/ Subject drops out due to logistic reasons and not due to any event related to treatment | <ul> <li>The strategy will be a While-on-Treatment strategy, where we are interested in the treatment effects prior to the withdrawal only.</li> <li>Subjects' data available up to the withdrawal will be included in the food effect analyses.</li> <li>If a subject withdraws consent during a period, the missing data post withdrawal will not be imputed.</li> <li>The derived PK parameters for e.g., AUC, C<sub>max</sub> etc. of that partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria).</li> </ul> |

| Subject does not take the full treatment | Not related to treatment/ The treatment will be administered as a powder dissolved in diluent. To ensure all treatment is ingested, the bottle containing the dispersion will be rinsed three times and the subject will be expected to ingest this in addition to the initial dispersion. If three rinses are not all ingested, the subject may not take the full treatment dose. | In the current formulation, it is hard to measure the exact proportion of dose ingested if not all rinses are taken. It is also uncertain whether the formulation could change in future development. To account for this, we propose two different strategies described below. If this intercurrent event is not observed, then both strategies will provide the same results and only the hypothetical strategy will be presented for the final analysis. Primary analysis - The strategy will be a Hypothetical strategy, where we are interested in the treatment effects in a hypothetical scenario where all subjects have taken complete dose. - In this case, the data from a period in which an incomplete dose is taken would be considered as missing at random and excluded from analyses. - If the drug formulation is changed in the future studies, this estimate will provide the true relationship between the actual dose intake and its exposure under this strategy. Supplementary analysis - The strategy will be a Treatment policy strategy, where we are interested in the treatment effects regardless of the actual amount of dose taken. - The analysis will include PK parameters derived based on concentrations of both complete and partial doses (if data permits based on criteria described in Section 8.1.1.2) and will be analysed using the nominal or prescribed dose |
|---|---|---|
| | | <ul> <li>and will be analysed using the nominal or prescribed dose.</li> <li>If the drug formulation remains unchanged in the future studies, this estimate will provide the true relationship between a nominal dose and its exposure under this strategy, i.e., close to a real-world situation.</li> </ul> |
| Subject<br>drops out<br>due to | Related to treatment/ If the adverse event is confirmed | - The primary strategy will be a <b>Hypothetical</b> strategy, where we are interested in the treatment effects in a hypothetical scenario where discontinuation due to an AE would not happen. |

| be related to udy treatment | - | The missing data after discontinuation will assumed to be missing at random The derived PK parameters of the last fully or partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |
|---|---|---|
|---|---|---|

## 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in ****: List of Data Displays and will be based on GSK Data Standards and statistical principles. Graphical presentations will be provided if appropriate. All data will be listed.

## 8.2.5.1. Statistical Methodology Specification

The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

## (1) Statistical analysis for comparison of food effect – Single dose study part

## **Endpoint / Variables**

- AUC (0-t)
- AUC(0-∞)
- Cmax

#### **Model Specification**

- Log<sub>e</sub>-transformed data will be statistically analysed using a Mixed model.
- The mixed model will contain
  - Fixed effect: fed or fasted status, period and their interaction term (if tested as significant)
  - o Random effect: subject
- Only data of subjects participating in Cohort 3 will be included in this analysis, all other dose level data from Cohorts 1 and 2 will be excluded from this analysis.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured type of the covariance matrices R (accounting for the within subject variability) and G (accounting for the between subject variability) will be used.
- Based on the intercurrent events observed in the study, appropriate strategies from Table 3
  in Section 8.2.4 will be considered for handling of missing data (if any) and interpretation of
  food effect analysis results. If multiple intercurrent events are observed (for e.g., if the

subject does not take the full treatment as well he withdraws study consent), then the data will be handled using more than one strategy as described in Table 3 and interpretations of the results will be made accordingly.

# **Model Checking & Diagnostics**

- For the Mixed model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold for any of the alternative transformations.
- If this model fails to converge, alternative covariance structures may be considered in the following order (1) Compound Symmetry (CS) and (2) Variance Components (VC).

#### **Model Results Presentation**

- Point estimates and corresponding 90% confidence intervals will be constructed for the comparisons of interest of GSK3186899 fed – GSK3186899 fasted, based on the logtransformed data.
- These loge-transformed results will then be exponentially back-transformed to provide point estimates and corresponding 90% confidence intervals for the geometric mean ratios (GSK3186899 fed: GSK3186899 fasted).

# 8.3. Statistical analysis for dose proportionality – Single and Repeat dose study parts

# 8.3.1. Endpoints/Variables

To assess the dose proportionality, the statistical analysis will be based on AUC, Cmax and Ctau variables, as appropriate in the single and repeat dose study part.

## 8.3.2. Summary Measure

The summary measure will be the point estimates and 90% CIs of mean slopes of log<sub>e</sub>(dose) in the single and repeat dose study part.

## 8.3.3. Population of Interest

These analyses will be based on the PK population.

## 8.3.4. Strategy for Intercurrent (Post-Randomization) Events

In the Table 4 below, the possible intercurrent events and the rationale for relating them to treatment or otherwise is described. Once a subject discontinues from study treatment, they will proceed straight to follow up and no further data will be collected.

All subjects' data will be included in data listings irrespective of the strategies followed for the analysis.

If feasible, subjects will be replaced until the desired sample size is attained.

**Table 4 Strategies for Intercurrent events** 

| Intercurrent events | Relation to treatment and rationale | Strategy, rationale and details of action taken |
|---|---|---|
| Subject<br>withdraws<br>study<br>consent | Not related to treatment/ Subject drops out due to logistic reasons and not due to any event related to treatment | <ul> <li>The strategy will be a While-on-Treatment strategy, where we are interested in the treatment effects prior to the withdrawal only.</li> <li>Subjects' data available up to the withdrawal will be included in the dose proportionality analyses.</li> <li>If a subject withdraws consent during a period, the missing data post withdrawal will not be imputed.</li> <li>The derived PK parameters for e.g., AUC, C<sub>max</sub> etc. of that partially completed period will be calculated if data permits (See section</li> </ul> |
| | | 8.1.1.2 Derived Pharmacokinetic Parameters |
|---|---|---|
| | | for details on derivation criteria). |
| Subject does not take the full treatment | Not related to treatment/ The treatment will be administered as a powder dissolved in diluent. To ensure all treatment is ingested, the bottle containing the dispersion will be rinsed three times and the subject will be expected to ingest this in addition to the initial dispersion. If three rinses are not all ingested, the subject may not take the full treatment dose. | In the current formulation, it is hard to measure the exact proportion of dose ingested if not all rinses are taken. It is also uncertain whether the formulation could change in future development. To account for this, we propose two different strategies described below. If this intercurrent event is not observed, then both strategies will provide the same results and only the hypothetical strategy will be presented for the final analysis. Primary analysis - The strategy will be a Hypothetical strategy, where we are interested in the treatment effects in a hypothetical scenario where all subjects have taken complete dose. - In this case, the data from a period in which an incomplete dose is taken would be considered as missing at random and excluded from analyses. - If the drug formulation is changed in the future studies, this estimate will provide the true relationship between the actual dose intake and its exposure under this strategy. Supplementary analysis - The strategy will be a Treatment policy strategy, where we are interested in the treatment effects regardless of the actual amount of dose taken. - The analysis will include PK parameters derived based on concentrations of both complete and partial doses (if data permits based on criteria described in Section 8.1.1.2) and will be analysed using the nominal or prescribed dose. - If the drug formulation remains unchanged in the future studies, this estimate will provide the true relationship between a nominal dose and its exposure under this strategy, i.e., in a close to real-world setting |
| Subject drops out | Related to treatment/ | - The primary strategy will be a <b>Hypothetical</b> strategy, where we are interested in the |

| due to<br>Adverse<br>events | If the adverse event is confirmed to be related to study treatment | - | treatment effects in a hypothetical scenario where discontinuation due to an AE would not happen. The missing data after discontinuation will assumed to be missing at random The derived PK parameters of the last fully or partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |
|---|---|---|---|
|---|---|---|---|

## 8.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in ****: List of Data Displays and will be based on GSK Data Standards and statistical principles. Graphical presentations will be provided if appropriate. All data will be listed.

## 8.3.5.1. Statistical Methodology Specification

The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

### (2) Statistical analysis for dose proportionality – Single and Repeat dose study parts

#### **Endpoint / Variables**

- For SAD part: AUC(0-∞), Cmax
- For MAD part: AUC(0-tau), Cmax, Ctau

## **Model Specification**

Power model

$$v = \alpha * dose^{\beta}$$

where y denotes the PK parameter being analyzed, dose denotes the total dose administered to a subject. The  $\alpha$  denotes random subject effect in the repeat dose Part B. In the crossover single ascending dose Part A, alpha depends upon random subject effect and period effect.

- Log<sub>e</sub> transformed data will be analysed by fitting the following terms in the mixed effect model:
  - Fixed effect: log<sub>e</sub> (dose), period (period will be included in SAD part only)
  - o Random effect: Subject
  - Data from all available doses in each part of the study will be considered (as described in Section 8.1.1.2).

- An unstructured covariance structure will be considered for the G matrix describing the between subject variability.
- Based on the intercurrent events observed in the study, appropriate strategies from
  Table 4 in Section 8.3.4 will be considered for handling of missing data (if any) and
  interpretation of the analysis results. If multiple intercurrent events are observed (for
  e.g., if the subject does not take the full treatment as well he withdraws study consent),
  then the data will be handled using more than one strategy as described in Table 4 and
  interpretations of the results will be made accordingly.

## **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined
  by obtaining a normal probability plot of the residuals and a plot of the residuals
  versus the fitted values (i.e., checking the normality assumption and constant
  variance assumption of the model respectively) to gain confidence that the model
  assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold for any of the alternative transformations.

#### **Model Results Presentation**

Estimates of the mean slopes of log<sub>e</sub>(dose) will be reported along with corresponding 90% confidence intervals (slope ≈ 1 implied dose proportionality).

# 8.4. Statistical analysis for dose accumulation – Repeat dose study part

## 8.4.1. Endpoints/Variables

To assess the dose accumulation, the statistical analysis will be based on the ratios of RAUC(0-tau), RCmax and RCtau respectively.

## 8.4.2. Summary Measure

The summary measure will be the point estimates and 90% CIs of mean differences of 'Day 10 - Day 1' based on the log-transformed data and after back-transformation of this estimated differences, the geometric means of the ratio 'Day 10: Day 1' will be presented.

## 8.4.3. Population of Interest

These analyses will be based on the PK population.

## 8.4.4. Strategy for Intercurrent (Post-Randomization) Events

In the Table 5 below, the possible intercurrent events and the rationale for relating them to treatment or otherwise is described. Once a subject discontinues from study treatment, they will proceed straight to follow up and no further data will be collected.

All subjects' data will be included in data listings irrespective of the strategies followed for the analysis.

If feasible, subjects will be replaced until the desired sample size is attained.

**Table 5 Strategies for Intercurrent events** 

| Intercurrent events | Relation to treatment and rationale | Strategy, rationale and details of action taken |
|---|---|---|
| Subject<br>withdraws<br>study<br>consent | Not related to treatment/ Subject drops out due to logistic reasons and not due to any event related to treatment | <ul> <li>The strategy will be a While-on-Treatment strategy, where we are interested in the treatment effects prior to the withdrawal only.</li> <li>Subjects' data available up to the withdrawal will be included in the dose accumulation analyses.</li> <li>If a subject withdraws consent during a period, the missing data post withdrawal will not be imputed.</li> <li>The derived PK parameters for e.g., AUC, Cmax etc. of that partially completed period will be calculated if data permits (See section</li> </ul> |

| | | 8.1.1.2 Derived Pharmacokinetic Parameters |
|---|---|---|
| | | for details on derivation criteria). |
| Subject does not take the full treatment | Not related to treatment/ The treatment will be administered as a powder dissolved in diluent. To ensure all treatment is ingested, the bottle containing the dispersion will be rinsed three times and the subject will be expected to ingest this in addition to the initial dispersion. If three rinses are not all ingested, the subject may not take the full treatment dose. | In the current formulation, it is hard to measure the exact proportion of dose ingested if not all rinses are taken. It is also uncertain whether the formulation could change in future development. To account for this, we propose two different strategies described below. If this intercurrent event is not observed, then both strategies will provide the same results and only the hypothetical strategy will be presented for the final analysis. Primary analysis - The strategy will be a Hypothetical strategy, where we are interested in the treatment effects in a hypothetical scenario where all subjects have taken complete dose. - In this case, the data from a period in which an incomplete dose is taken would be considered as missing at random and excluded from analyses. - If the drug formulation is changed in the future studies, this estimate will provide the true relationship between the actual dose intake and its exposure under this strategy. Supplementary analysis - The strategy will be a Treatment policy strategy, where we are interested in the treatment effects regardless of the actual amount of dose taken. - The analysis will include PK parameters derived based on concentrations of both complete and partial doses (if data permits based on criteria described in Section 8.1.1.2) and will be analysed using the nominal or prescribed dose. - If the drug formulation remains unchanged in the future studies, this estimate will provide the true relationship between a nominal dose and its exposure under this strategy, i.e., close to a real-world setting. |
| Subject drops out | Related to treatment/ | - The primary strategy will be a <b>Hypothetical strategy</b> , where we are interested in the |

| due to<br>Adverse<br>events | If the adverse event is confirmed to be related to study treatment | - | treatment effects in a hypothetical scenario where discontinuation due to an AE would not happen. The missing data after discontinuation will assumed to be missing at random The derived PK parameters of the last fully or partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |
|---|---|---|---|
|---|---|---|---|

## 8.4.5. Statistical Analyses / Methods

Details of the planned displays are provided in ****: List of Data Displays and will be based on GSK Data Standards and statistical principles. Graphical presentations will be provided if appropriate. All data will be listed.

## 8.4.5.1. Statistical Methodology Specification

The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

### Statistical analysis for dose accumulation – Repeat dose study part

#### **Endpoint / Variables**

- RAUC(0-tau)
- RCmax
- RCtau

### **Model Specification**

- Will be statistically analysed using a mixed model (MM) using a log<sub>e</sub>-transformation. The mixed model will contain:
  - Fixed effects: dose, day and dose\*day
  - o Random effect: Subject

Here dose denotes the total dose administered per day to a subject.

- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured type of the covariance matrices R (accounting for the within subject variability) and G (accounting for the between subject variability) will be used.
- Based on the intercurrent events observed in the study, appropriate strategies from Table 5
  in Section 8.4.4 will be considered for handling of missing data (if any) and interpretation of
  the analysis results. If multiple intercurrent events are observed (for e.g., if the subject does

not take the full treatment as well he withdraws study consent), then the data will be handled using more than one strategy as described in Table 5 and interpretations of the results will be made accordingly.

## **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold for any of the alternative transformations.
- If this model fails to converge, alternative covariance structures may be considered in the following order (1) Compound Symmetry (CS) and (2) Variance Components (VC).

#### **Model Results Presentation**

- For each dose, point estimates and 90% confidence intervals for the differences "Day 10 -Day 1" will be presented based on the log-transformed data.
- These point estimates and associated 90% confidence intervals will then be exponentially back-transformed to provide point and 90% confidence interval estimates for the ratios "Day 10: Day 1" for each active dose.
- If both the dose and day by dose interaction terms are not significant, and only day effect is significant based on the data, then to evaluate the effect of day, a single point estimate and confidence interval pooled across all doses by day will be constructed.

# 8.5. Statistical analysis for time invariance ratio of GSK3186899 - Repeat dose study part

## 8.5.1. Endpoints/Variables

To assess the time invariance dose accumulation, the statistical analysis will be based on the ratio of AUC(0-tau) (i.e., AUC(0-12) if dosing is BID or, AUC(0-8) if dosing is TID) on day 10 to AUC(0- $\infty$ ) on day 1, if data permits.

## 8.5.2. Summary Measure

The summary measure will be the point estimate and 90% CIs of mean difference of 'AUC(0-tau) at Day  $10 - \text{AUC}(0-\infty)$  at Day 1' based on the log-transformed data and after back-transformation of this estimated difference, the geometric mean of the ratio 'AUC(0-tau) at Day 10 : AUC(0- $\infty$ ) at Day 1' will also be presented.

## 8.5.3. Population of Interest

This analysis will be based on the PK population.

## 8.5.4. Strategy for Intercurrent (Post-Randomization) Events

In the Table 6 below, the possible intercurrent events and the rationale for relating them to treatment or otherwise is described. Once a subject discontinues from study treatment, they will proceed straight to follow up and no further data will be collected.

All subjects' data will be included in data listings irrespective of the strategies followed for the analysis.

If feasible, subjects will be replaced until the desired sample size is attained.

**Table 6 Strategies for Intercurrent events** 

| Intercurrent events | Relation to treatment and rationale | Strategy, rationale and details of action taken |
|---|---|---|
| Subject<br>withdraws<br>study<br>consent | Not related to treatment/ Subject drops out due to logistic reasons and not due to any event related to treatment | <ul> <li>The strategy will be a While-on-Treatment strategy, where we are interested in the treatment effects prior to the withdrawal only.</li> <li>Subjects' data available up to the withdrawal will be included in the time invariance accumulation rate analyses.</li> <li>If a subject withdraws consent during a period, the missing data post withdrawal will not be imputed.</li> <li>The derived PK parameters for e.g., AUC, Cmax etc. of that partially completed period</li> </ul> |

| | | will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |
|---|---|---|
| Subject does not take the full treatment | Not related to treatment/ The treatment will be administered as a powder dissolved in diluent. To ensure all treatment is ingested, the bottle containing the dispersion will be rinsed three times and the subject will be expected to ingest this in addition to the initial dispersion. If three rinses are not all ingested, the subject may not take the full treatment dose. | In the current formulation, it is hard to measure the exact proportion of dose ingested if not all rinses are taken. It is also uncertain whether the formulation could change in future development. To account for this, we propose two different strategies described below. If this intercurrent event is not observed, then both strategies will provide the same results and only the hypothetical strategy will be presented for the final analysis. Primary analysis - The strategy will be a Hypothetical strategy, where we are interested in the treatment effects in a hypothetical scenario where all subjects have taken complete dose. - In this case, the data from a period in which an incomplete dose is taken would be considered as missing at random and excluded from analyses. - If the drug formulation is changed in the future studies, this estimate will provide the true relationship between the actual dose intake and its exposure under this strategy. Supplementary analysis - The strategy will be a Treatment policy strategy, where we are interested in the treatment effects regardless of the actual amount of dose taken. - The analysis will include PK parameters derived based on concentrations of both complete and partial doses (if data permits based on criteria described in Section 8.1.1.2) and will be analysed using the nominal or prescribed dose. - If the drug formulation remains unchanged in the future studies, this estimate will provide the true relationship between a nominal dose and its exposure under this strategy, i.e. close to a real-world setting. |

| Subject<br>drops out<br>due to<br>Adverse<br>events | Related to treatment/ If the adverse event is confirmed to be related to study treatment | - | The primary strategy will be a <b>Hypothetical strategy</b> , where we are interested in the treatment effects in a hypothetical scenario where discontinuation due to an AE would not happen. The missing data after discontinuation will assumed to be missing at random The derived PK parameters of the last fully or partially completed period will be calculated if data permits (See section 8.1.1.2 Derived Pharmacokinetic Parameters for details on derivation criteria). |
|---|---|---|---|
|---|---|---|---|

## 8.5.5. Statistical Analyses / Methods

Details of the planned displays are provided in ****: List of Data Displays and will be based on GSK Data Standards and statistical principles. Graphical presentations will be provided if appropriate. All data will be listed.

## 8.5.5.1. Statistical Methodology Specification

The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

## Statistical analysis for time invariance ratio of GSK3186899 – Repeat dose study part

#### **Endpoint / Variables**

Ratio of AUC(0-tau) on day 10 to AUC(0-∞) on day 1

(This will be calculated only if  $AUC(0-\infty)$  on day 1 is appropriately estimated)

#### **Model Specification**

- Will be statistically analysed using a mixed model (MM) using a log<sub>e</sub>-transformation. The mixed model will contain:
  - Fixed effects: day
  - o Random effect: Subject
- AUC(0-∞) on day 1 will be the reference phase in the analysis, while AUC(0-tau) on day 10 will be the test phase for BID (or, TID) regimen respectively, using loge-transformed AUC.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured type of the covariance matrices G (accounting for the between subject variability) will be used.

Based on the intercurrent events observed in the study, appropriate strategies from Table 6 in Section 8.5.4 will be considered for handling of missing data (if any) and interpretation of the analysis results. If multiple intercurrent events are observed (for e.g., if the subject does not take the full treatment as well he withdraws study consent), then the data will be handled using more than one strategy as described in Table 6 and interpretations of the results will be made accordingly.

## **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined
  by obtaining a normal probability plot of the residuals and a plot of the residuals
  versus the fitted values (i.e. checking the normality assumption and constant
  variance assumption of the model respectively) to gain confidence that the model
  assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold for any of the alternative transformations.
- If this model fails to converge, alternative covariance structures may be considered in the following order (1) Compound Symmetry (CS) and (2) Variance Components (VC).

### **Model Results Presentation**

• The summary measure will be the point estimate and 90% CIs of mean difference of 'AUC(0-tau) at Day 10 – AUC(0-∞) at Day 1' based on the log-transformed data and after back-transformation of this estimated difference, the geometric mean of the ratio 'AUC(0-tau) at Day 10 : AUC(0-∞) at Day 1' will also be presented.

## 9. REFERENCES

- Alves F, Bilbe G, Blesson S et al. Recent development of visceral leishmaniasis treatments: success, pitfalls and perspectives. *Clin Microbiol Rev.* 2018 Aug 29; 31(4):e00048-18.
- Committee for Human Medicinal Products. ICH E9 (R1) addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials, Step 2b. London: European Medicines Evaluation Agency, August 2017.
- Dorlo TP, Rijal S, Ostyn B, de Vries PJ, Singh R, Bhattarai N, Uranw S, Dujardin JC, Boelaert M, Beijnen JH, Huitema AD. Failure of miltefosine in visceral leishmaniasis is associated with low drug exposure. *J Infect Dis.* 2014 Jul 1;210(1):146-53.
- Dorlo TP1, Huitema AD, Beijnen JH, de Vries PJ. Optimal dosing of miltefosine in children and adults with visceral leishmaniasis. *Antimicrob Agents Chemother*. 2012 Jul;56(7):3864-72.
- FDA Guidance for industry: Estimating the maximum safe dose in initial clinical trials for therapeutics in adult healthy volunteers. 2005 <a href="http://www.fda.gov/downloads/Drugs/Guidances/UCM078932.pdf">http://www.fda.gov/downloads/Drugs/Guidances/UCM078932.pdf</a>

## 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 10.1.1. Exclusions from Analysis Population

Per protocol population is not defined in this protocol.

Important protocol deviations and violations of the inclusion and exclusion criteria will be listed.

# 10.2. Appendix 2: Schedule of Activities

## 10.2.1. Protocol Defined Schedule of Events in PART A (Cohorts 1-3)

| | Screening | S | tudy F | eriod | (Days | s) | Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -1 | 1 | 2 | 3 | 4 | (14-21 days post<br>last dose)<br>/Early<br>Withdrawal | Notes |
| Outpatient Visit | X | | | | | | Χ | |
| Admission to Clinical Unit | | Χ | | | | | | |
| Inpatient Stay at Clinical Unit | | <b>←</b> | ==== | ==X== | ==== | | | |
| Discharge from Clinical Unit | | | | | | Χ | | Following completion of all assessments. |
| Informed Consent | X | | | | | | | |
| Inclusion and Exclusion Criteria | X | | | | | | | |
| Demography | X | | | | | | | |
| Full Physical Examination | Х | | | | | | | Additional exams/screens may be performed, or brief exams made full exams, by the Investigator, as deemed necessary (e.g. where safety or laboratory findings indicate). Tests will be conducted within site |
| Brief Physical Examination | | Χ | | Χ | | Χ | X | specified standards. |
| Drug/Alcohol/Smoking Screen | X | Χ | | | | | | Tests include alcohol breath test, smoking breath test and urine drug screen. |
| Medical/Medication/Drug/Alcohol<br>History | Х | | | | | | | |
| HIV, Hepatitis B and C Screening | Х | | | | | | | |
| FSH + Oestradiol | Х | | | | | | | Females only, if required |
| Holter Monitoring (48 hours) | Х | | | | | | | |
| Haem/Chem/Urinalysis Test<br>(Include Liver Chemistries) | х | Х | | Х | | Х | Х | If trace protein in urine is detected, a repeat test can be performed (within 24 hours). If tests are considered abnormal, further quantification is required. |
| | | | | | | | | Non-fasted samples can be collected on Day -1 and the Follow-Up Visit. All other samples to be collected in a fasted state. |
| Urine Sampling (metabolism) | | | Х | Х | | | | A urine sample will be taken pre-dose (approx. 20mL) All urine from each participant will be collected from 0-24 hrs post dosing. Details of urine collection and processing are described in the SRM. |

| | Screening | Study Period (Days) | | | | | Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -1 | 1 | 2 | 3 | 4 | (14-21 days post<br>last dose)<br>/Early<br>Withdrawal | Notes |
| Safety biomarkers (KIM1, NGAL,<br>Urinary albumin) | | | Х | х | | | | First urine sample of the morning to be collected (Day 1 sample collection should be pre-dose). Additional samples may be collected, as deemed necessary by the Investigator (e.g. where safety or laboratory findings indicate). |
| PK Blood Sampling | | | Х | х | | | | PK blood samples to be taken pre-dose on Day 1 and then at the following time points post first-dose: 10min, 30min, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 5hr, 6hr, 8hr, 10hr, 12hr; 24hr. The time points stated may be modified depending on emerging SAD PK information as appropriate. Blood volumes to be collected include 2 mL for all time-points from pre-dose to 10 hrs, and 5 mL for time-points 12hr and 24 hr. |
| 12-Lead ECG | Х | Χ | Т | Х | <b>←</b> > | $\langle \rightarrow$ | | Vital signs to include HR, BP, temperature and respiration rate. BP will be conducted in both a supine and standing position if participant |
| Vital Signs | X | x | Т | x | <b>←</b> > | <del>(→</del> | X | develops any signs/symptoms which in the investigator's opinion are suggestive of adrenal insufficiency. 12-Lead ECG and Vital Signs to be conducted on Day -1 and pre-dose on Day 1 and then at the subsequent time points post-dose: 30 min, 1 hr, 1.5hr, 2hr, 2.5hr, 4hr, 8hs, 12hr, 24 hr, 48 hr Timings will be reviewed as cohorts progress and may be adjusted to ensure appropriate measurements relative to peak concentrations for subsequent cohorts. T = Triplicate (for all assessments, except temperature and respiratory rate). If any abnormal ECG reading is recorded, refer to Section Error! Reference source not found. for appropriate action. |

| | Screening | St | tudy F | Period | (Days | 5) | Follow-Up | |
|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -1 | 1 | 2 | 3 | 4 | (14-21 days post<br>last dose)<br>/Early<br>Withdrawal | Notes |
| Telemetry | | | <b>←</b> > | ⟨→ | | | | Continuous at least 24hr post-dose. Initiate at least 15 min. prior to dosing. |
| Meals | | Х | X | X | X | X | | Fasting regimen: On Day 1, participants will have fasted 8hr overnight prior to dosing. An adapted standard breakfast will be served approximately 3 hours after dosing. Fed regimen: On Day 1, participants will fast 8hr overnight and an adapted standard breakfast will be served approximately 30 minutes prior to dosing. Meals will be served as per the site schedule on Days -1, 2, 3 and 4. Water permitted on an ad lib basis up to 1hr before dosing. No water to be taken in the hour prior to dosing except for the liquid part of the adapted standard breakfast for the Fed regimen. At least 8 fl oz (240ml) to be taken 1 hour after dosing. No water to be taken in the hour after dosing except for the dose. |
| Bile Sampling (Entero-test) | | | Χ | | | | | <b>Cohort 3 only.</b> Entero-test bile string swallowed 2 hr post-dose, after 5 hr the bile string will be removed. |
| Randomization | | | Χ | | | | | |
| Study Treatment | | | Χ | | | | | |
| AE Review | | | | ==X== | | | X | |
| SAE Review | X | • | | ==X== | | | X | |
| Concomitant Medication Review | Х | ←= | ==== | ==X== | ==== | <del>-</del> → | X | |

# 10.2.2. Protocol Defined Schedule of Events in PART B (Cohorts 4-6)

| | Screening | | | | | | S | tudy | Perio | d (Day | rs) | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| Outpatient Visit | Х | | | | | | | | | | | | | | | | Х | |
| Admission to Clinical Unit | | Х | | | | | | | | | | | | | | | | |
| Inpatient Stay at<br>Clinical Unit | | | • | <del>(</del> === | ==== | ==== | ==== | ==== | ====) | X===: | | ==== | ==== | ==== | ====- | <del>)</del> | | |
| Discharge from<br>Clinical Unit | | | | | | | | | | | | | | | | Х | | Following completion of all assessments. |
| Informed Consent | Χ | | | | | | | | | | | | | | | | | |
| Inclusion and Exclusion Criteria | Х | | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | | |
| Full Physical<br>Examination | Х | | | | | | | | | | | | | | | | | Additional exams/screens may be performed, or brief exams made full |
| Brief Physical<br>Examination | | | Х | | x | | | | | X | | | | | | х | X | exams, by the Investigator, as deemed necessary (e.g. where safety or laboratory findings indicate). Tests will be conducted within site specified standards. |
| Drug/Alcohol/Smoki<br>ng Screen | Х | | Х | | | | | | | | | | | | | | | Tests include alcohol breath test, smoking breath test and urine drug screen. |
| Medical/Medication/<br>Drug/Alcohol<br>History | Х | | | | | | | | | | | | | | | | | |
| HIV, Hepatitis B and C Screening | Х | | | | | | | | | | | | | | | | | |
| FSH + Oestradiol | X | | | | | | | | | | | | | | | | | Females only, if required |
| Holter Monitoring (48 hour) | Х | | | | | | | | | | | | | | | | | |

| | Screening | | | | | | S | Study | Perio | d (Day | /s) | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| Haem/Chem/<br>Urinalysis Test<br>(Include Liver<br>Chemistries) | X | | X | | X | | X | | X | | X | | X | | X | X | X | If trace protein is detected, a repeat test can be performed. Sample to be drawn pre-dose on Days 2, 4, 6, 8 and 10. Non-fasted samples can be collected on Day -1 and Follow-Up Visit. All other samples to be collected in fasted state. |
| Cortisol Test | | | Х | | | | | | | | | | | x | | | | Tests to be performed in the early morning on Day -1 and Day 11. If levels are <420 nmol/L, then a ACTH stimulation test will be performed to assess hypothalamic pituitary adrenal (HPA) axis. |
| Safety biomarkers<br>(KIM1, NGAL,<br>Urinary albumin) | | | | X | | | | х | | | | | | | | | | First urine sample of the morning to be collected (pre-dose). Additional samples may be collected, as deemed necessary by the Investigator (e.g. where safety or laboratory findings indicate). |
| Telemetry | | | | X | Х | | | | | | | | | | | | | Continuous at least 24 hr post-evening dose. Initiate at least 15 min. prior to dosing. |
| Randomization | | | | Χ | | | | | | | | | | | | | | |
| Study Treatment | | | | Х | Х | Χ | х | Х | х | х | Χ | х | Χ | | | | | BID dosing: GSK3186899 or placebo will be administered using a 12hr dosing interval. If a different dosing regimen is used, refer to Appendix 5 of Protocol. |

| | Screening | | | | | | S | Study | Perio | d (Day | /s) | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| 12-Lead ECG | Х | | Х | Т | Х | | Х | | Х | | Х | | Х | | Х | Х | X | Vital signs to include HR, BP, temperature and respiration rate. BP will be conducted in both a supine and standing position if participant develops any signs/symptoms |
| Vital signs | X | | X | Т | X | X | X | Х | X | X | X | X | X | X | X | X | X | which in the investigators opinion are suggestive of adrenal insufficiency. 12-Lead ECG and Vital Signs to be conducted on Day-1 and pre-dose Day 1 and then at the subsequent time points post first-dose: 30 min, 1 hr, 1.5hr, 2hr, 2.5hr, 4hr, 6hr, 13hr and 14hr For Days 2-10: pre-dose assessments only. Timings will be reviewed as cohorts progress and may be adjusted to ensure appropriate measurements relative to peak concentrations for subsequent cohorts If a different dosing regimen is used, refer to Appendix 5 for alternative ECG and Vital Signs time-points. T = Triplicate (for all assessments except temperature and respiratory rate). If any abnormal ECG reading is recorded, refer to Section Error! Reference source |

| | Screening | | | | | | S | Study | Perio | d (Day | rs) | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| | | | | | | | | | | | | | | | | | | <b>not found.</b> of protocol for appropriate action. |
| PK Blood sampling | | | | <== | | ====: | | | ==X== | | | | ====: | ==> | | | | PK samples will be collected pre-dose and at the following time points post first-dose: Day 1: 10min, 30min, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 5hr, 6hr, 8hr, 10hr, and 12hr Days 2 – 9: Pre-dose PK samples collected for each dose Day 10: PK samples will be collected pre-dose and at the following time points post first-dose: 10min, 30min, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 5hr, 6hr, 8hr, 10hr, and 12hr. The time points stated may be modified depending on emerging SAD PK profiles. If a different dosing regimen is used, refer to Appendix 5 of Protocol for alternative PK blood sampling time-points. Blood volumes to be collected include: 2 mL for post-dose 0-11 hrs, and 5 mL for post-dose 12-24 hrs (Days 1 and 10). |
| Urine Sampling<br>(metabolism) | | | | | | | | | | | | | Х | X | | | | A urine sample will be taken pre-dose (approx. 20mL). All urine from each participant will be collected from 0-24 hrs post dosing. Details of urine collection and processing are described in the SRM. |

| | Screening | | | | | | S | Study | Perio | d (Day | /s) | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| Meals AE review | | X | X | X | X | X | X | X | X<br>==X=: | X | X | X | X | X | X | X | X | If on fed regimen: On Day 1 through to D10, participants will receive an adapted standard meal 30 mins prior to dosing. If on fasted regimen: On Day 1 through to D10, participants will have fasted 8hr overnight prior to dose 1. A breakfast will be served approximately 2hr after dose 1. Dinner will be served at least 2hr prior to dose 2. A snack may be consumed approximately 2hr after dose 2. Participants will receive standardized meals scheduled at the same time in each period. If a different dosing regimen is used, refer to Appendix 5 for alternative meal times. Meals will be served as per the site schedule on Days -1 and Days 11-13. Water permitted on an ad lib basis up to 1hr before dosing. No water to be taken in the hour prior to dosing except for the liquid part of the adapted standard breakfast for the Fed regimen. At least 8 fl oz (240ml) to be taken 1 hour after dosing No water to be taken in the hour after dosing except for the rinse of the dose. |

| | Screening | | Study Period (Days) | | | | | | | | | | | | | | Follow-up<br>(14-21 days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (Up to 28<br>days before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | post last<br>dose) /<br>Early<br>Withdrawal | Notes |
| SAE review | Х | + | -=== | ==== | ==== | | ==== | | :==X=: | ==== | ==== | ==== | ==== | ==== | ==== | $\rightarrow$ | Х | |
| Concomitant medication review | Х | + | -=== | ==== | ==== | | ==== | | ==X= | | ==== | ==== | | ==== | ==== | · <b>→</b> | Х | |

• The timing and number of planned study assessments, including safety, pharmacokinetic or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/IEC will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the informed consent form (ICF).

## 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Assessment Windows for Analyses

Nominal time will be used for all analysis except PK analysis where planned and actual time will be used.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 10.4.1. Study Phases

For each period in Part A Cohorts 1, 2 and 3, assessments and events will be classified according to the following phases:

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date and time < Study Treatment Start Date and time of each period |
| Treatment | Study Treatment Start Date and time ≤ Date and time ≤ Study Treatment End Date and time + 24 hours, in each period |
| Post-Treatment | Date and time > Study Treatment End Date and time + 24 hours, within each period |

Note: Estimated half-life of GSK3186899 is approx. 1.3 hours. The maximum of (5 half-lives (~ 6.5 hours) and 24 hours) after the Study Treatment End Date and time have been considered to define the end of treatment phase. If half-life is longer than 5 hours, then the definition will be revised accordingly.

Post-treatment phase will additionally include any events occurring in the washout period before start of the next treatment dose.

For the interim, the start of the period will be defined from the first dose of the period and then the end of the period is just before the first dose in the next period. For the final period the end date is just before the withdrawal/follow up visit.

For Part B Cohorts 4, 5 and 6, assessments and events will be classified according to the following:

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date of each Cohort |
| Treatment | Study Treatment Start Date and time ≤ Date and time ≤ Study Treatment End Date and time + 24 hours, in each cohort |
| Post-Treatment | Date and time > Study Treatment End Date and time 24 hours, in each cohort |

Note: Estimated half-life of GSK3186899 is approx. 1.3 hours. The maximum of (5 half-lives (~ 6.5 hours) and 24 hours) after the Study Treatment End Date and time have been considered to define the end of treatment phase. If half-life is longer than 5 hours, then the definition will be revised accordingly.

#### 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before to the screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment Emergent | If AE onset date is on or after treatment start date and time, it is considered as treatment emergent |
| | • For Part A, if AE onset is during one period and worsens during a later period it would be counted in both periods. |
| | <ul> <li>For the initial period the logic would be as above.</li> </ul> |
| | <ul> <li>For the later period the logic would use the treatment dates<br/>associated with the later period:</li> </ul> |
| | Treatment Period Start Date ≤ AE Worsening Date ≤ Study<br>Treatment Stop Date |

### NOTES:

- If the study treatment stop date is missing, then the AE will be considered as On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently support to the currently su | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | :\\UK1SALX00175.corpnet2.com\ |
| HARP Compound | : \arprod\gsk3186899\mid208436\ |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1] | |
| Generation of RTF Files | |
| RTF files will be generated for SAC. | |

## 10.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles as indicated below but may be adjusted to a clinically interpretable number of DP's.
  - Display all numeric variables with the same number of decimal places as the collected precision.
  - Display minimum and maximum values with the same number of decimal places as the collected precision.
  - Display the mean and percentiles (e.g. median, Q1, and Q3) with one additional decimal place.
  - Display the standard deviation and standard error with two additional decimal places.
  - Within a column, align all data values or summary statistics along the decimal point.

The reported precision for PK concentration data will be 1 decimal place but may be altered by parameter depending on the significant digits.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and figures.
- All unscheduled visits will be included in listings.

| | <b>5</b> |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | orical Data N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [SOP_514512]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | None. All PK parameters will be derived by the CPMS Pharmacokineticist. |
| Pharmacokinetic Para | nmeter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters guidance. |
| Descriptive Summary<br>Statistics, Graphical | Refer to IDSL PK Display Standards. |
| Displays and Listings | Log <sub>e</sub> -transformed data: |
| | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of loge transformed data and between subject |

## CONFIDENTIAL

208436

geometric coefficient of variation (CV<sub>b</sub> (%)) will be reported. CV<sub>b</sub> (%) =  $\sqrt{(exp(SD^2) - 1) * 100}$  [NOTE: SD = SD of log<sub>e</sub> transformed data]

Parameters Not Being Log\_e Transformed: Tmax and T1/2.

## 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day and Period Study Day

- In PART A for each period: Period Study day is calculated as the number of days from first Dose Date in the period for each subject as follows:
  - Ref Date = Missing → Period Study Day = Missing
  - Ref Date < First Dose Date in the period → Period Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date in the period → Period Study Day = Ref Date First Dose Date + 1
- In Part A and Part B: Study day is calculated as the number of days from First Dose Date in each Cohort for each subject as:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 10.6.2. Study Population

#### **Treatment Exposure and Compliance**

#### For Parts A and B:

Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Doses taken/ (Planned Treatment Duration in Days \* Frequency)

where Frequency will be 1 for OD, 2 for BID or 3 for TID. Treatment compliance could be greater than 100% if there are events of overdose.

- Planned Treatment Duration is defined as 10 days, for each Cohort in Part B. As Part A is single dose this would be one day.
- Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure (in Days) = Treatment Stop Date - (Treatment Start Date) + 1

 Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

#### For Part B:

• The cumulative dose will be based on the formula:

**Cumulative Dose = Sum of (Number of Days x Total Daily Dose)** 

#### **Treatment Exposure and Compliance**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

## Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

## 10.6.3. Safety

#### **Adverse Events**

#### [AE'S OF Special Interest]

- Stomach erosion
- Adrenal insufficiency
- Renal impairment (Note: Protocol defines renal stopping and withdrawal criteria which are not "renal impairment" in the strict sense)

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places = '< x' becomes x 0.01
  - Example 2: 1 Decimal Places = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places = '< x' becomes x 1
  - o For values '<=x' or '>=x' the value itself ('x') should be imputed as the numeric value.
- Renal biomarker data will be included in the final study analysis. The parameters will be corrected using the following formula, and the units are ng/mg
   Corrected KIM-1=8.8\*Urine KIM-1(pG/mL)/Urine Creatinine (umol/L)
   Corrected NGAL=8800\*Urine NGAL(nG/mL)/Urine Creatinine (umol/L)

#### 10.6.4. Pharmacokinetic

### PK parameters

- The PK Population will include all subjects who undergo PK sampling and have evaluable PK concentration results.
- See Section 8.1 for derived Pharmacokinetic parameters

# 10.7. Appendix 7: Reporting Standards for Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as the completion of all phases of the study including the last scheduled procedure shown in SoA (Appendix 2). The end of study is defined as the date of the last visit of the last participant in the study or last scheduled procedure shown in the SoA for the last participant in the trial.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. Unless specified otherwise,</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> <li>Missing safety data (for e.g., lab, ECG, Vitals, etc.) will not be imputed.</li> <li>Missing PK data may be imputed (if required) by the Estimand strategy and will be outlined in the final RAP.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | Missing or Partial start/end date and time are not expected for Adverse events. |
| Concomitant<br>Medications/<br>Medical<br>History | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: • If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month • If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. The recorded partial date will be displayed in listings. • For assigning periods: |

## CONFIDENTIAL

| Element | Reporting Detail |
|---|---|
| | If start date is completely missing, then we assume the medication has been taken from the beginning of the study |
| | <ul> <li>If stop date is completely missing, then we assume the medication has been taken<br/>until the end of the study</li> </ul> |
| | If start and stop date are completely missing, then we assume the medication has been |
| | taken for the duration of the study |

# 10.8. Appendix 8: Values of Potential Clinical Importance

The values of potential clinical importance for Laboratory, ECG and Vital signs are listed in this section.

## 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | <37 | >50 |
| Hematocrit | % | Female | <33 | >45 |
| | | $\Delta$ from BL | N/A | > 7.5% |
| | /1 | Male | <130 | >170 |
| Hemoglobin | g/L | Female | <115 | >155 |
| | | $\Delta$ from BL | N/A | > 30 g/L |
| Lymphocytes | x10 <sup>9</sup> / L | | <1.2 | >3.65 |
| Neutrophils | x10 <sup>9</sup> / L | | <2 | >7.5 |
| Monocytes | x10 <sup>9</sup> / L | | <0.2 | >1 |
| Basophils | x10 <sup>9</sup> / L | | <0.0 | >0.1 |
| Platelet Count | x10 <sup>9</sup> / L | | <150 | >400 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | <3.0 | >10 |
| Red Blood Cell Count (RBC) | x10 <sup>12</sup> /L | Male | <4.4 | >5.8 |
| - 133 2.333 33.: 30an (1.23) | | Female | <3.95 | >5.15 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | < 34 | > 50 |
| Calcium | mmol/L | | < 2.2 | > 2.6 |
| Creatinine | umol/L | Male | < 66 | > 112 |
| Creatifile | ullioi/L | Female | < 49 | > 92 |
| Glucose (Fasted) | mmol/L | | < 3.9 | > 5.8 |
| Magnesium | mmol/L | | < .6 | >1 |
| Phosphate | mmol/L | | < 0.87 | > 1.45 |
| Potassium | mmol/L | | < 3.5 | > 5.1 |
| Sodium | mmol/L | | < 135 | > 145 |
| Gamma GT | g/L | | < 7.7 | > 17.3 |

| Liver Function | | | | |
|---|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Alkalina phaanhataaa | U/L | Female | < 35 | > 104 |
| Alkaline phosphatase | U/L | Male | < 40 | > 129 |
| AST/SGOT | U/L | Male | < 0 | > 37 |
| A31/3G01 | U/L | Female | < 0 | > 31 |
| ALT/SGPT | U/L | Male | < 10 | > 50 |
| AL1/SGP1 | U/L | Female | < 10 | > 35 |
| Total Bilirubin | µmol/L | | < 0 | > 20 |
| Direct Bilirubin | µmol/L | | < 0 | > 20 |
| Total Protein | g/L | | < 63 | > 83 |

## 10.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTcF during the | msec | | >500 |
| study (i.e. post dose) | | | |
| Absolute PR Interval | msec | < 110 | >220 |
| Absolute QRS Interval | msec | < 75 | >120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |
| Tympanic temperature | °C | <35 | >38 |
| Respiratory rate | Breaths/min | <10 | >25 |

# 10.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Not applicable.

# 10.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

Not applicable.

## 10.11. Appendix 11: Abbreviations & Trade Marks

## 10.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| AUC | Area under the concentration-time curve |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DEC | Dose escalation committee |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FTIH | First Time in Human |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |

| Abbreviation | Description 208436 |
|--------------|----------------------------------------------------------|
| IP | Investigational Product |
| LDH | · · |
| MAD | Lactate Dehydrogenase |
| | Multiple Ascending Dose |
| MCH | Mean Corpuscular Haemoglobin |
| MCV | Mean Corpuscular Volume |
| NGAL | Neutrophil gelatinase-associated lipocalin |
| NOAEL | No Observable Adverse Effect Limit |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTc | Electrocardiogram QT interval corrected for heart rate |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RBC | Red Blood Cells |
| RAUC | Relative Area Under the Curve |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAD | Single Ascending dose |
| SAE | Serious Adverse Event |
| SDD | Spray Dried Dispersion |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SGOT | Serum Glutamic-Oxaloacetic Transaminase |
| SGPT | Serum Glutamic-Pyruvic Transaminase |
| SOA | Schedule of Activities |
| SOP | Standard Operation Procedure |
| SRM | Study Reference Manual |
| SUSAR | Suspected Unexpected Serious Adverse Events |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TID | Three-Times Daily |
| Tmax | Time Taken to Maximum Observed Plasma Drug Concentration |
| | Lag time before observation of drug concentrations |
| Tlag<br>t1/2 | Terminal phase half-life |
| τ | Dosing interval |
| UK | United Kingdom |
| ULN | Upper Limit of Normal |
| VL | Visceral Leishmaniasis |
#### CONFIDENTIAL

208436

| Abbreviation | Description |
|--------------|--------------------------------------|
| WONCBP | Women of Non-Child Bearing Potential |

## 10.11.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |
| NONMEM |

## 10.12. Appendix 12: List of Data Displays

### 10.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|----------------|----------------|
| Study Population | 1.1 to 1.22 | None |
| Efficacy | Not applicable | Not applicable |
| Safety | 3.1 to 3.34 | None |
| Pharmacokinetic | 4.1 to 4.11 | 4.1 to 4.10 |
| Section | Listings | |
| ICH Listings | 1 to 65 | |
| Other Listings | 66 to 80 | |

### 10.12.2. Mock Example Shell Referencing

Non-integrated data standards library (IDSL) specifications will be referenced as indicated and if required example mock-up displays provided in

Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' column as '[Non-Standard] + Reference.'

#### 10.12.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------------------------|
| IA | Informal Interim Analysis (displays to be prepared by |
| | Biostatistics function) |
| SAC | Final Statistical Analysis Complete |

# 10.12.4. Study Population Tables

| Study Po | pulation Tab | es | | | |
|---|---|---|---|---|---|
| No. | Populati on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Subject [ | Disposition | | | • | |
| 1.1. | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record – Part A | ICH E3, FDAAA, EudraCT | IA, SAC |
| 1.2. | Safety | ES1 | Summary of Participant Disposition for the Participant Conclusion Record – Part B | ICH E3, FDAAA, EudraCT | SAC |
| 1.3. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment – Part B | ICH E3 | SAC |
| 1.4. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part A | ICH E3 | SAC |
| 1.5. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part B | ICH E3 | SAC |
| 1.6. | Screene<br>d | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part A | | SAC |
| 1.7. | Screene<br>d | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part B | | SAC |
| Protocol | Deviation | | | | |
| 1.8. | Safety | DV1 | Summary of Important Protocol Deviations – Part A | ICH E3 | SAC |
| 1.9. | Safety | DV1 | Summary of Important Protocol Deviations – Part B | ICH E3 | SAC |
| Population | on Analysed | | | | |
| 1.10. | Enrolled | SP1 | Summary of Study Populations – Part A | | IA, SAC |
| | • | | | | |

| Study Po | pulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.11. | Enrolled | SP1 | Summary of Study Populations – Part B | | SAC |
| Demogra | phic and Bas | eline Characteris | tics | | |
| 1.12. | Safety | DM3 | Summary of Demographic Characteristics – Part A | ICH E3, FDAAA, EudraCT | IA, SAC |
| 1.13. | Safety | DM1 | Summary of Demographic Characteristics – Part B | ICH E3, FDAAA, EudraCT | SAC |
| 1.14. | Enrolled | DM11 | Summary of Age Ranges – Part A | EudraCT | SAC |
| 1.15. | Enrolled | DM11 | Summary of Age Ranges – Part B | EudraCT | SAC |
| 1.16. | Safety | DM5 | Summary of Race and Racial Combinations – Part A | ICH E3, FDA, FDAAA, EudraCT | SAC |
| 1.17. | Safety | DM5 | Summary of Race and Racial Combinations – Part B | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Prior and | l Concomitan | t Medications | | | • |
| 1.18. | Safety | CM1 | Summary of Concomitant Medications – Part A | ICH E3 | SAC |
| 1.19. | Safety | CM1 | Summary of Concomitant Medications – Part B | ICH E3 | SAC |
| Exposure | and Treatmen | t Compliance | | | |
| 1.20. | Safety | EX1 | Summary of Exposure to Study Treatment – Part A | ICH E3 | IA, SAC |
| 1.21. | Safety | EX1 | Summary of Exposure to Study Treatment - Part B | ICH E3 | SAC |
| 1.22. | Safety | COMP1 | Summary of Overall Compliance Based on Exposure –Part B | | SAC |

# 10.12.5. Safety Tables

| Safety: Tal | bles | | | | |
|---|---|---|---|---|---|
| No. | Populat ion | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Adverse E | vents (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term – Part A | ICH E3 | IA, SAC |
| 3.2. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term – Part B | ICH E3 | SAC |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part A | FDAAA, EudraCT | SAC |
| 3.4. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part B | FDAAA, EudraCT | SAC |
| 3.5. | Safety | AE1 | Summary of All Drug Related Adverse Events by System Organ Class and Preferred Term – Part A | ICH E3 | SAC |
| 3.6. | Safety | AE1 | Summary of All Drug Related Adverse Events by System Organ Class and Preferred Term – Part B | ICH E3 | SAC |
| Serious an | nd Other Sig | nificant Adverse l | Events | | |
| 3.7. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Part A | FDAAA, EudraCT | SAC |
| 3.8. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Part B | FDAAA, EudraCT | SAC |
| Laboratory | y: Chemistr | у | | | |
| 3.9. | Safety | LB1 | Summary of Chemistry Changes from Baseline – Part A | ICH E3 | SAC |
| 3.10. | Safety | LB1 | Summary of Chemistry Changes from Baseline – Part B | ICH E3 | SAC |

| Safety: Ta | bles | | | | |
|---|---|---|---|---|---|
| No. | Populat ion | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.11. | Safety | LB17 | Summary of Worst-Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline – Part A | ICH E3 | SAC |
| 3.12. | Safety | LB17 | Summary of Worst-Case Chemistry Results by PCI Criteria<br>Post-Baseline Relative to Baseline – Part B | ICH E3 | SAC |
| Laborator | y: Haematol | ogy | | 1 | |
| 3.13. | Safety | LB1 | Summary of Haematology Changes from Baseline – Part A | ICH E3 | SAC |
| 3.14. | Safety | LB1 | Summary of Haematology Changes from Baseline – Part B | ICH E3 | SAC |
| 3.15. | Safety | LB17 | Summary of Worst-Case Haematology by PCI Criteria Post-<br>Baseline Relative to Baseline – Part A | ICH E3 | SAC |
| 3.16. | Safety | LB17 | Summary of Worst-Case Haematology by PCI Criteria Post-<br>Baseline Relative to Baseline – Part B | ICH E3 | SAC |
| Laborator | y: Urinalysi | S | | 1 | |
| 3.17. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline – Part A | ICH E3<br>Includes Baseline values. | SAC |
| 3.18. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline – Part B | ICH E3<br>Includes Baseline values. | SAC |
| 3.19. | Safety | UR3a | Summary of Urinalysis Dipstick and Microscopy Results – Part A | | SAC |
| 3.20. | Safety | UR3a | Summary of Urinalysis Dipstick and Microscopy Results – Part B | | SAC |
| 3.21. | Safety | UR1 | Summary of Worst-Case Urinalysis Results Post-Baseline Relative to Baseline – Part A | ICH E3 | SAC |
| 3.22. | Safety | UR1 | Summary of Worst-Case Urinalysis Results Post-Baseline Relative to Baseline – Part B | ICH E3 | SAC |
| Laborator | y: Hepatobi | liary (Liver) | | | |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Populat ion | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.23. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part A | | SAC |
| 3.24. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part B | | SAC |
| 3.25. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities – Part A | | SAC |
| 3.26. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities – Part B | | SAC |
| ECG | | | | | |
| 3.27. | Safety | EG1 | Summary of ECG Findings – Part A | | SAC |
| 3.28. | Safety | EG1 | Summary of ECG Findings – Part B | | SAC |
| 3.29. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit – Part A | Includes Baseline values. | SAC |
| 3.30. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit – Part B | Includes Baseline values. | SAC |
| Vital Sign | S | 1 | | 1 | <u> </u> |
| 3.31. | Safety | VS1 | Summary of Change from Baseline in Vital Signs - Part A | ICH E3 Includes Baseline values. | SAC |
| 3.32. | Safety | VS1 | Summary of Change from Baseline in Vital Signs - Part B | ICH E3 Includes Baseline values. | SAC |
| 3.33. | Safety | VS7 | Summary of Worst-Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline – Part A | | SAC |
| 3.34. | Safety | VS7 | Summary of Worst-Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline – Part B | | SAC |

#### 10.12.6. Pharmacokinetic Tables

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Pharm | acokinetic Con | centration Data | | | |
| 4.1. | PK | PK01 | Summary of GSK3186899 Plasma Pharmacokinetic Concentration-Time Data - Part A | | SAC |
| 4.2. | PK | PK01 | Summary of GSK3186899 Plasma Pharmacokinetic Concentration-Time Data - Part B | | SAC |
| Derive | d Pharmacokin | etic Parameters | | | |
| 4.3. | PK | PK06 | Summary of Non-transformed Derived GSK3186899 Plasma Pharmacokinetic Parameters by Dose - Part A | | SAC |
| 4.4. | PK | PK06 | Summary of Non-transformed Derived GSK3186899 Plasma<br>Pharmacokinetic Parameters by Dose - Part B | | SAC |
| 4.5. | PK | PK05 | Summary of Log <sub>e</sub> -Transformed Derived GSK3186899 Plasma<br>Pharmacokinetic Parameters by Dose - Part A | | SAC |
| 4.6. | PK | PK05 | Summary of Loge-Transformed Derived GSK3186899 Plasma<br>Pharmacokinetic Parameters by Dose - Part B | | SAC |
| 4.7. | PK | Non-standard<br>PK_T1 | Statistical analysis for comparison of food effect in Part A Cohort 3 | | SAC |
| 4.8. | PK | Non-standard<br>PK_T2 | Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part A | | SAC |
| 4.9. | PK | Non-standard<br>PK_T3 | Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part B | | SAC |
| 4.10. | PK | Non-standard<br>PK_T4 | Statistical Analysis of Log-transformed Plasma GSK3186899<br>Parameters Assessing Steady-State – Part B | | SAC |

| P | Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. Population IDSL / Example Shell Title Programming Notes | | | | Deliverable | | |
| 4 | .11. | PK | Non-standard<br>PK_T4 | Time invariance analysis of log-transformed Plasma<br>GSK3186899 Parameters – Part B | Update the parameters for time invariance analysis | SAC |

# 10.12.7. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Pharma | Pharmacokinetic Concentration Data | | | | |
| 4.1. | PK | PK16 | Individual Plasma GSK3186899 Concentration-Time Plot (Linear and Semi-Log)– Part A | | SAC |
| 4.2. | PK | PK16 | Individual Plasma GSK3186899 Concentration-Time Plot (Linear and Semi-Log)– Part B | | SAC |
| 4.3. | PK | PK19 | Mean (+ SD) Plasma GSK3186899 Concentration-Time Plots (Linear and Semi-Log)- Part A | | SAC |
| 4.4. | PK | PK19 | Mean (+ SD) Plasma GSK3186899 Concentration-Time Plots (Linear and Semi-Log)- Part B | | SAC |
| 4.5. | PK | PK20 | Median (range) Plasma GSK3186899 Concentration-Time Plots (Linear and Semi-Log)- Part A | | SAC |
| 4.6. | PK | PK20 | Median (range) Plasma GSK3186899 Concentration-Time Plots (Linear and Semi-Log)- Part B | | SAC |
| Derive | d Pharmacokin | etic Parameters | | | |
| 4.7. | PK | Non-standard<br>PK_F1 | Box Plot of AUC(0-∞) and Cmax versus dose (Linear) – Part A | | SAC |
| 4.8. | PK | Non-standard<br>PK_F1 | Box Plot of AUC(0-∞) and Cmax versus dose (Linear) – Part B | AUC(0-tau) on day 10 | SAC |
| 4.9. | PK | Non-standard<br>PK_F1 | Box Plot of dose normalised AUC(0-∞) versus dose (Linear) – Part A | | SAC |
| 4.10. | PK | Non-standard<br>PK_F1 | Box Plot of dose normalised AUC(0-∞) and Cmax versus dose (Linear) - Part B | AUC(0-tau) on day 10 | SAC |

# 10.12.8. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure – Part A | | SAC |
| 2. | Screened | ES7 | Listing of Reasons for Screen Failure – Part B | | SAC |
| 3. | Screened | ES9 | Listing of Subjects Who Were Rescreened by Cohort – Part A | | SAC |
| 4. | Screened | ES9 | Listing of Subjects Who Were Rescreened in Part B by Cohort – Part B | | SAC |
| 5. | Safety | ES3 | Listing of Reasons for Study Withdrawal – Part A | ICH E3 | IA, SAC |
| 6. | Safety | ES2 | Listing of Reasons for Study Withdrawal – Part B | ICH E3 | SAC |
| 7. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation – Part A | ICH E3 | IA, SAC |
| 8. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation – Part B | ICH E3 | SAC |
| 9. | Enrolled | BL1 | Listing of Participants for Whom the Treatment Blind was Broken – Part A | ICH E3 | SAC |
| 10. | Enrolled | BL1 | Listing of Participants for Whom the Treatment Blind was Broken – Part B | ICH E3 | SAC |
| 11. | Enrolled | TA1 | Listing of Planned and Actual Treatments - Part A | | SAC |
| 12. | Enrolled | TA1 | Listing of Planned and Actual Treatments - Part B | | SAC |
| Protoc | ol Deviations | | | | |
| 13. | Safety | DV2 | Listing of Important Protocol Deviations – Part A | ICH E3 | IA, SAC |
| 14. | Safety | DV2 | Listing of Important Protocol Deviations – Part B | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 15. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations - Part A | ICH E3 | SAC |
| 16. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations – Part B | ICH E3 | SAC |
| Popula | tions Analysed | I | | | • |
| 17. | Safety | SP3 | Listing of Subjects Excluded from Any Population – Part A | ICH E3 | SAC |
| 18. | Safety | SP3 | Listing of Subjects Excluded from Any Population – Part B | ICH E3 | SAC |
| Demog | raphic and Bas | seline Characteris | etics | | |
| 19. | Safety | DM4 | Listing of Demographic Characteristics – Part A | ICH E3 Include BMI and smoking status. | IA, SAC |
| 20. | Safety | DM2 | Listing of Demographic Characteristics – Part B | ICH E3 Include BMI and smoking status. | SAC |
| 21. | Safety | DM9 | Listing of Race – Part A | ICH E3 | SAC |
| 22. | Safety | DM9 | Listing of Race – Part B | ICH E3 | SAC |
| Prior a | nd Concomitar | nt Medications | | | • |
| 23. | Safety | CP_CM3 | Listing of Concomitant Medications- Part A | IDSL | SAC |
| 24. | Safety | CP_CM3 | Listing of Concomitant Medications- Part B | IDSL | SAC |
| Expos | ure and Treatm | ent Compliance | | | • |
| 25. | Safety | EX4 | Listing of Exposure Data - Part A | ICH E3 | IA, SAC |
| 26. | Safety | EX3 | Listing of Exposure Data - Part B ICH E3 | | SAC |
| 27. | Safety | COMP2 | Listing of Compliance Based on Exposure –Part B | | |
| Advers | se Events | | | | |
| 28. | Safety | AE9 | Listing of All Adverse Events – Part A | ICH E3 | IA, SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 29. | Safety | AE8 | Listing of All Adverse Events – Part B | ICH E3 | SAC |
| 30. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events – Part A | ICH E3 | SAC |
| 31. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events – Part B | ICH E3 | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 32. | Safety | AE8CP | Listing of Serious Adverse Events – Part A | ICH E3 | SAC |
| 33. | Safety | AE8CP | Listing of Serious Adverse Events – Part B | ICH E3 | SAC |
| 34. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse<br>Event- Part A | ICH E3 | SAC |
| 35. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse<br>Event- Part B | ICH E3 | SAC |
| 36. | Safety | AECP8 | Listing of Adverse Events Leading to Withdrawal from Study – Part A | ICH E3 | SAC |
| 37. | Safety | AECP8 | Listing of Adverse Events Leading to Withdrawal from Study – Part B | ICH E3 | SAC |
| 38. | Safety | AECP8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment – Part A | ICH E3 | SAC |
| 39. | Safety | AECP8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment – Part B | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | |
| 40. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events - Part A | IDSL | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Listing of Medical Conditions for Subjects with Liver Stopping | | Title | Programming Notes | Deliverable |
| 41. | | | IDSL | SAC | |
| 42. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events - Part A | IDSL | SAC |
| 43. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events - Part B | IDSL | SAC |
| All Lab | oratory | | | | , |
| 44. | Safety | of Potential Clinical Importance – Part A subject who experienced a | | ICH E3 Display ALL chemistry data for a subject who experienced a value of potential clinical importance. | IA, SAC |
| 45. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance – Part B | ICH E3 Display ALL chemistry data for a subject who experienced a value of potential clinical importance. | SAC |
| 46. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance – Part A | | SAC |
| 47. | Safety | LB5 | Listing of Laboratory Values of Potential Clinical Importance – Part B | | SAC |
| 48. | Safety | LB14 | Listing of Laboratory Data with Character Results – Part A | ICH E3 | SAC |
| 49. | Safety | LB14 | Listing of Laboratory Data with Character Results – Part B | ICH E3 | SAC |
| 50. | Safety UR2B Listing of All Urinalysis Data for Subjects with Any Value of Potential Clinical Importance – Part A | | ICH E3 Display ALL urinalysis data for a subject who experienced a value of potential clinical importance. | IA, SAC | |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title | | Title | Programming Notes | Deliverable |
| 51. | Safety | UR2A | Listing of All Urinalysis Data for Subjects with Any Value of Potential Clinical Importance – Part B ICH E3 Display ALL urinalysis data fo subject who experienced a value of potential clinical importance. | | SAC |
| 52. | Safety | UR2B | Listing of Urine Biomarker data for all Subjects – Part A | Only present urine biomarker data | SAC |
| 53. | Safety | UR2A | Listing of Urine Biomarker data for all Subjects – Part B | Only present urine biomarker data | SAC |
| ECG | | | | | |
| 54. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance – Part A | IDSL Display ALL ECG data for a subject who experienced a value of potential clinical importance. | IA, SAC |
| 55. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance – Part B | IDSL Display ALL ECG data for a subject who experienced a value of potential clinical importance. | SAC |
| 56. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance – Part A | IDSL | SAC |
| 57. | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance – Part B | IDSL | SAC |
| 58. | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding – Part A | | IA, SAC |
| 59. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding – Part B | IDSL | SAC |
| Vital Sig | gns | | | | |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 60. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance – Part A | IDSL Display ALL vital signs data for a subject who experienced a value of potential clinical importance. | IA, SAC |
| 61. | Safety | VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance – Part B | IDSL Display ALL vital signs data for a subject who experienced a value of potential clinical importance. | SAC |
| 62. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance – Part A | IDSL | SAC |
| 63. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance – Part B | IDSL | SAC |
| 64. | Safety | EG6 | Listing of Telemetry findings - Part A | Example shell to be modified for telemetry data | IA, SAC |
| 65. | Safety | EG5 | Listing of Telemetry findings - Part B | Example shell to be modified for telemetry data | SAC |

# 10.12.9. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Safety | | | | | |
| 66. | Safety | HM10 | Listing of Clinically Significant Holter Abnormalities – Part A | | SAC |
| 67. | Safety | HM10 | Listing of Clinically Significant Holter Abnormalities – Part B | | SAC |
| 68. | Safety | МН3 | Listing of Medical conditions – Part A | | SAC |
| 69. | Safety | MH2 | Listing of Medical conditions – Part B | | SAC |
| Pharm | acokinetic | | | | |
| 70. | PK | PK07 | Listing of Plasma GSK3186899 Pharmacokinetic Concentration-Time Data – Part A | | SAC |
| 71. | PK | PK07 | Listing of Plasma GSK3186899 Pharmacokinetic Concentration-Time Data – Part B | | SAC |
| 72. | PK | PK13 | Listing of Derived Plasma GSK3186899 Pharmacokinetic Parameters – Part A | | SAC |
| 73. | PK | PK13 | Listing of Derived Plasma GSK3186899 Pharmacokinetic Parameters – Part B | | SAC |
| 74. | PK | PK07 | PK07 Listing of Urine GSK3186899 Pharmacokinetic Concentration-Time Data – Part A Only include 3 Urine PK parameters: Ae(t1-tz), fe(0-tz), CLR | | SAC |
| 75. | PK | PK07 | Listing of Urine GSK3186899 Pharmacokinetic Concentration-Time Data – Part B | Only include 3 Urine PK parameters:<br>Ae(t1-tz), fe(0-tz), CLR | SAC |
| 76. | PK | Non-standard | Raw SAS output of Statistical Analysis for Comparison of Food effect - Part A Cohort 3 | | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title | | Title | Programming Notes | Deliverable |
| 77. | PK | Non-standard | Raw SAS output of Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part A | | SAC |
| 78. | PK | Non-standard | Raw SAS output of Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part B | | SAC |
| 79. | PK | Non-standard | Raw SAS output of Statistical Analysis of Log-transformed Plasma GSK3186899 Parameters Assessing Steady-State – Part B | | SAC |
| 80. | PK | Non-standard | Raw SAS output of Time invariance analysis of log-<br>transformed Plasma GSK3186899 Parameters – Part B | | SAC |

### 10.13. Appendix 13: Example Mock Shells for Data Displays

Example : PK T1

Population : Pharmacokinetic

| Parameter Fed (Units) | | Fa | sted | GSK X.X mg Fed vs Fasted (Difference) | 90% CI of<br>the<br>difference | GSK X.X<br>mg<br>Fed vs<br>Fasted<br>(Ratio) | 90% CI<br>of the<br>Ratio | |
|---|---|---|---|---|---|---|---|---|
| | n | LS Mean | n | LS Mean | | | | |
| AUC(0-t) (µg.h/mL) | Х | XX.XX | Х | XX.XX | x.xx | (x.xx,<br>x.xx) | x.xx | (x.xx,<br>x.xx) |
| Cmax<br>(µg/mL) | Х | xx.xx | Х | xx.xx | x.xx | (x.xx,<br>x.xx) | x.xx | (x.xx,<br>x.xx) |

Log-transformed parameter is modelled with fed or fasted status and period as fixed effects and subject as a random effect. Unstructured covariance structures are considered describing within and between subject variability.

A ratio of 1 indicates same PK response is seen in both the fed and fasted subjects. A ratio > 1 indicates a higher PK response was seen in the fed subjects.

Example : PK T2

Population : Pharmacokinetic

Table 4.8

Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) - Part A

| Parameter (Units) | Slope | 90% CI of the Slope |
|---|---|---|
| | Log Parameter vs Log Dose | |
| <auc(0-t) (µg.h="" ml)=""></auc(0-t)> | X.XX | (x.xx, x.xx) |
| Cmax (µg/mL) | X.XX | (x.xx, x.xx) |

A Power model is used to assess the dose proportionality.

 $Log_e$  (dose) and period are fitted as fixed effects and subject as a random effect. An unstructured covariance structure is considered describing between subject variability.

A slope of 1 indicates the pharmacokinetics are dose proportional. A slope greater than 1 indicates the increase in PK is greater than proportional to dose.

Example : PK T3

Population : Pharmacokinetic

Table 4.9

Statistical Analysis of Log Transformed Plasma GSK3186899 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) - Part B

| Parameter (Units) | Timepoint | Slope | 90% CI of the |
|---|---|---|---|
| | | Log Parameter vs Log Dose | Slope |
| <auc(0-t) (µg.h="" ml)=""></auc(0-t)> | Day 1 | x.xx | (x.xx, x.xx) |
| | Day 10 | X.XX | (x.xx, x.xx) |
| Cmax (µg/mL) | Day 1 | X.XX | (x.xx, x.xx) |
| | Day 10 | X.XX | (x.xx, x.xx) |
| | · | | |

A Power model is used to assess the dose proportionality.

 $Log_e$  (dose) is fitted as a fixed effect and subject as a random effect. An unstructured covariance structure is considered describing between subject variability.

A slope of 1 indicates the pharmacokinetics are dose proportional. A slope greater than 1 indicates the increase in PK is greater than proportional to dose.

Example : PK T4

Population : Pharmacokinetic

Table 4.10

Statistical Analysis of Log Transformed Plasma GSK3186899 Trough Concentration Assessing Steady-State - Part B

| Parameter | Treatment | Day 10 | | Day 1 | | Log- | 90% | Back- | 90% |
|---|---|---|---|---|---|---|---|---|---|
| (Units) | | _ | | | | transformed | Confidence | Transformed | Confidence |
| | | | | | | Day 10 - | Interval | Ratios | Interval |
| | | | | | | Day 1 | | | |
| | | n | LS | n | LS Mean | | | | |
| | | | Mean | | | | | | |
| Ctau | <dose 1=""></dose> | X | XX.XX | X | XX.XX | X.XX | (x.xx, | X.XX | (x.xx, |
| (ug/mL) | | | | | | | x.xx) | | x.xx) |
| | <dose 2=""></dose> | Х | XX.XX | Х | XX.XX | X.XX | (x.xx, | X.XX | (x.xx, |
| | | | | | | | x.xx) | | x.xx) |
| | <dose 3=""></dose> | Х | XX.XX | Х | XX.XX | X.XX | (x.xx, | X.XX | (x.xx, |
| | | | | | | | x.xx) | | x.xx) |

A Mixed effect model including dose, day and dose-by-day interaction as fixed effects and subject as a random effect is used to assess accumulation ratios. Unstructured covariance structures are used to describe within and between subject variabilities. A ratio of 1 indicates no accumulation. A ratio > 1 indicates drug accumulation.

Example : PK\_F1

Population: Pharmacokinetic

Figure 4.7
Box Plot of AUC and Cmax versus doses (Linear) - Part A



Period 2 60 mg
Period 3 120 mg

Programming notes: this is an example shell to be updated to present each dose level.